# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population Phase II

Protocol CR-6267

Version: 2.0 Amendment 1

Date: 22 June 2018

Investigational Products: JJV Investigational senofilcon A Multifocal Contact Lens and 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens

Key Words: Presbyopia, Multifocal, etafilcon A, senofilcon A, Daily Wear, Daily Disposable, Reusable, Dispensing, Randomized

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

# **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# TABLE OF CONTENTS

| PROTO | OCOL TITLE, NUMBER, VERSION | 6 |
|---|---|---|
| | SOR NAME AND ADDRESS | |
| | CAL MONITOR | |
| | ORIZED SIGNATURES | |
| | GE HISTORY | |
| | PSIS | |
| | IONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | |
| | TRODUCTION AND BACKGROUND | |
| 1.1. | Name and Descriptions of Investigational Products | |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | |
| 1.5. | Relevant Literature References and Prior Clinical Data Relevant to | |
| Clini | cal Study | |
| 2. ST | TUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 18 |
| 2.1. | Objectives | 18 |
| 2.2. | Endpoints | 18 |
| 2.3. | Hypotheses | 18 |
| 3. TA | ARGETED STUDY POPULATION | 19 |
| 3.1. | General Characteristics | 19 |
| 3.2. | Inclusion Criteria | 19 |
| 3.3. | Exclusion Criteria | 19 |
| 3.4. | Enrollment Strategy | 20 |
| 4. ST | TUDY DESIGN AND RATIONALE | 20 |
| 4.1. | Description of Study Design | 20 |
| 4.2. | Study Design Rationale | 20 |
| 4.3. | Enrollment Target and Study Duration | 21 |
| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 21 |
| 5.1. | Test Article Allocation | 21 |
| 5.2. | Masking | 21 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 22 |
| 6 ST | TIDY INTERVENTION | 22 |

| | 6.1. | Identity of Test Articles | 22 |
|----|--------|--------------------------------------------------|----|
| | 6.2 Aı | ncillary Supplies/Products | 23 |
| | 6.3. | Administration of Test Articles | 23 |
| | 6.4. | Packaging and Labeling | 23 |
| | 6.5. | Storage Conditions | 24 |
| | 6.6. | Collection and Storage of Samples | 24 |
| | 6.7. | Accountability of Test Articles | 24 |
| 7. | STU | JDY EVALUATIONS | 25 |
| | 7.1. | Time and Event Schedule | 25 |
| | 7.2. | Detailed Study Procedures | 29 |
| | VIS | SIT 1 | 29 |
| | VIS | SIT 2 | 35 |
| | VIS | SIT 3 | 39 |
| | VIS | SIT 4 | 44 |
| | VIS | SIT 5 | 50 |
| | VIS | SIT 6 | 55 |
| | VIS | SIT 7 | 59 |
| | FIN | AL EVALUATION | 62 |
| | 7.3. | Unscheduled Visits | 62 |
| | 7.4. | Laboratory Procedures | 64 |
| 8. | SU | BJECTS COMPLETION/WITHDRAWAL | 64 |
| | 8.1. | Completion Criteria | 64 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 64 |
| 9. | PR1 | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 65 |
| 1( | ). D | EVIATIONS FROM THE PROTOCOL | 65 |
| 1 | 1. S' | TUDY TERMINATION | 65 |
| 12 | 2. P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 66 |
| 13 | 3. A | DVERSE EVENTS | 67 |
| | 13.1. | Definitions and Classifications | 67 |
| | 13.2. | Assessing Adverse Events | 70 |
| | 13.2 | 2.1. Causality Assessment | 70 |
| | 13.2 | 2.2. Severity Assessment | 70 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 71 |
| | 13.4 | Reporting Adverse Events | 72 |

| | 13.4.1 | Reporting Adverse Events to Sponsor | 72 |
|---|---|---|---|
| | 13.4.2<br>Autho | 2. Reporting Adverse Events to the Responsible IEC/IRB and H | |
| | 13.4.3 | 3. Event of Special Interest | 73 |
| 13 | .5. | Reporting of Pregnancy | 73 |
| 14. | STA | ATISTICAL METHODS | 74 |
| 14 | .1. | General Considerations. | 74 |
| 14 | .2. | Sample Size Justification | 74 |
| 14 | .3. | Analysis Populations | 74 |
| 14 | .4. | Level of Statistical Significance | 75 |
| 14 | .5. | Primary Analysis | 75 |
| 14 | .6. | Secondary Analysis | 75 |
| 14 | .7. | Other Exploratory Analyses | 75 |
| 14 | .8. | Interim Analysis | 76 |
| 14 | .9. | Procedure for Handling Missing Data and Drop-Outs | 76 |
| 14 | .10. | Procedure for Reporting Deviations from Statistical Plan | 76 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 76 |
| 15 | .1. | Electronic Case Report Form/Data Collection | 76 |
| 15 | .2. | Subject Record | 77 |
| 16. | DA | TA MANAGEMENT | 77 |
| 16 | .1. | Access to Source Data/Document | 77 |
| 16 | .2. | Confidentiality of Information | 77 |
| 16 | .3. | Data Quality Assurance | 78 |
| 17. | MO | NITORING | 78 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 78 |
| 18 | .1. | Study-Specific Design Considerations | 78 |
| 18 | .2. | Investigator Responsibility | 79 |
| 18 | .3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 79 |
| 18 | .4. | Informed Consent | 80 |
| 18 | .5. | Privacy of Personal Data | 81 |
| 19. | STU | JDY RECORD RETENTION | 81 |
| 20. | | ANCIAL CONSIDERATIONS | |
| 21. | | BLICATION | |
| 22. | REI | FERENCES | 83 |
| APPI | ENDI | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 84 |

| APPENDIX B : PATIENT INSTRUCTION GUIDE | . 116 |
|-------------------------------------------------------------|-------|
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | . 117 |
| APPENDIX D: BINOCULAR OVER REFRACTION | |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | . 149 |
| APPENDIX F: OCULAR DOMINANCE | . 150 |
| APPENDIX G: Test LENS FITTING GUIDE | . 151 |
| APPENDIX H: CONTROL LENS FITTING GUIDE | . 153 |
| APPENDIX I: CLINICAL TECHNICAL PROCEDURES (CTP) | . 155 |
| LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS | . 156 |
| EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | |
| DETERMINATION OF NEAR ADDITION | . 169 |
| NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE | . 177 |
| LENS FITTING CHARACTERISTICS | . 180 |
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | . 187 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRI REFRACTIONS | |
| BIOMICROSCOPY SCALE | |
| KERATOMETRY PROCEDURE | |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCED | |
| DISTANCE LOGWAR VISUAL ACUITI MEASUREMENT PROCED | |
| Visual Acuity Chart Luminance and Room Illumination Testing | . 213 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | . 218 |
| TABLE OF CONTENTS | 12 |
| Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | 23 |
| Table 3: Time and Events | |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic

Population Phase II

Protocol Number: CR-6267 Version: 2.0 Amendment 1

Date: 22 June 2018

# **SPONSOR NAME AND ADDRESS**

Johnson & Johnson Vision (JJV) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**

Name: Thomas R. Karkkainen, OD, MS, FAAO

Title: Sr. Principal Research Optometrist

Address: 7500 Centurion Parkway, Jacksonville, Florida 32256

Email: TKarkkai@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### AUTHORIZED SIGNATURES

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Report | |
|---|---|---|
| | Thomas R. Karkkainen, OD, MS, FAAO<br>Sr. Principal Research Optometrist | DATE |
| Clinical Operations<br>Manager | See Electronic Signature Report | |
| | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | |
| | | DATE |
| Data Management | See Electronic Signature Report | |
| | | DATE |
| Reviewer | _See Electronic Signature Report | |
| | | DATE |
| Approver | See Electronic Signature Report | DATE |
| | | DATE |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| | | Number(s) Affected | |
| 1.0 | Tom | Original Protocol | 30-Apr-2018 |
| | Karkkainen | _ | _ |
| 2.0 | Tom | -Revised Section 6.1 Test Article the | 22-Jun-2018 |
| Amendment 1 | Karkkainen | Investigational Multifocal Lens Codes | |
| | | -Updated Version and Date throughout | |
| | | the Document. | |

# **SYNOPSIS**

| D 4 1 T'41 | |
|---|---|
| Protocol Title | Clinical Evaluation of a Reusable Multifocal Optical Design in |
| | a Presbyopic Population Phase II |
| Sponsor | JJV, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development phase, Phase 2 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Product: JJV Investigational Multifocal |
| | Contact Lens manufactured in senofilcon A material. |
| | Marketed Product: 1-Day Acuvue® Moist Brand Multifocal |
| | Contact Lens. |
| Wear and Replacement | Wear Schedule: The Test and Control lenses are used as daily |
| Schedules | wear (note: the Test lens will be reusable and the Control lens |
| Somedares | daily disposable). |
| | daily disposacio). |
| | Replacement Schedule: The Test lens will be replaced at the |
| | optimization visit. The Control lens will be replaced after |
| | each day of wear as well as the optimization visit and the visit |
| | after the first week of wear in the optimized pair. The Test |
| | and Control lenses will also be replaced when lost or damaged. |
| Ohioatiyas | |
| Objectives | This study is an evaluation of the visual performance, |
| | subjective response, lens fit and ocular physiological response |
| | of the JJV Investigational senofilcon A Multifocal Contact |
| | Lens. The Test lens will be compared to the 1-Day Acuvue® |
| | Moist Brand Multifocal Contact Lens manufactured in |
| | etafilcon A material for CLUE subjective vision. |
| Study Endpoints | Primary endpoints: CLUE vision scores |
| | Other observations: logMAR visual acuity scores, lens fit, |
| | summary of number of lenses needed to fit (optimize) the |
| | subject, CLUE comfort/handling scores, corneal staining, and |
| | ocular redness. |
| Study Design | This is a single-masked, randomized-controlled, dispensing |
| | clinical trial. A total of approximately 60 eligible hyperopic |
| | subjects will be targeted to complete the study. The subjects |
| | will be fit in each study lens and wear the lens for 2-4 days |
| | then undergo optimization, if applicable, and wear the |
| | optimized pair for approximately 2 weeks with a follow-up at |
| | 1 week. The primary endpoints will be CLUE vision scores. |
| Sample Size | A total of approximately 60 subjects will be targeted to |
| 1 | complete. |
| Study Duration | The study will last approximately 2-4 months. |
| 2.5.4) 2 41401011 | 1 222 222 37 THE INDU APPEARMENT IN 1 HIGHERTON |

| Anticipated Study | Healthy male and female volunteers with presbyopia will be |
|---|---|
| Population | invited to participate in the study. Subjects will be adapted |
| - | soft contact lens wearers in both eyes. Additional information |
| | regarding the eligibility of the population can be found in the |
| | inclusion/exclusion criteria outlined below. |
| Eligibility Criteria | Potential subjects must satisfy all the following criteria to be |
| | enrolled in the study |
| | 1. The subject must read, understand, and sign the |
| | STATEMENT OF INFORMED CONSENT and |
| | receive a fully executed copy of the form. |
| | 2. The subject must appear able and willing to adhere to |
| | the instructions set forth in this clinical protocol. |
| | 3. The subject must be between 40 and 70 years of age (inclusive). |
| | 4. The subject's distance spherical equivalent refraction |
| | must be in the range of +1.25 D to +3.75 D in each |
| | eye. |
| | 5. The subject's refractive cylinder must be ≤0.75 D in each eye. |
| | 6. The subject's ADD power must be in the range of |
| | +0.75 D to +2.50 D. |
| | 7. The subject must have best corrected visual acuity of |
| | 20/20 <sup>-3</sup> or better in each eye. |
| | 8. Subjects must own a wearable pair of spectacles if |
| | required for their distance vision. |
| | 9. The subject must be an adapted soft contact lens |
| | wearer in both eyes (i.e. worn lenses a minimum of 2 |
| | days per week for at least 8 hours per wear day, for 1 |
| | month of more duration). |
| | 10. The subject must either already be wearing a |
| | presbyopic contact lens correction (e.g., reading |
| | spectacles over contact lenses, multifocal or |
| | monovision contact lenses, etc.) or if not respond |
| | positively to at least one symptom on the "Presbyopic |
| | Symptoms Questionnaire". |
| | Potential subjects who meet any of the following criteria will |
| | be excluded from participating in the study: |
| | 1. Currently pregnant or lactating. |
| | 2. Any active or ongoing ocular or systemic allergies that |
| | may interfere with contact lens wear. |
| | 3. Any active or ongoing systemic disease, autoimmune |
| | disease, or use of medication, which may interfere with |
| | contact lens wear. This may include, but not be limited |
| | to, diabetes, hyperthyroidism, Sjögren's syndrome, |
| | xerophthalmia, acne rosacea, Stevens-Johnson |

| Medications/Interventions Measurements and Procedures | contact lens wear. 5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions. 6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.). 7. A history of amblyopia, strabismus or binocular vision abnormality. 8. Any current ocular infection or inflammation. 9. Any current ocular abnormality that may interfere with contact lens wear. 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids. 11. Use of any ocular medication, with the exception of rewetting drops. 12. History of herpetic keratitis. 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment. 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician). 15. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multi-purpose care solution or Eye-Cept® rewetting drop solution. Use of any prescription or over-the-counter (OTC) medications that may affect contact lens wear. See Section 7.2 for the detailed procedures. |
|---|---|
| Microbiology or Other Laboratory Testing | None |

| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
|---|---|
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, will result in stopping further dispensing |
| | investigational product. In the event of a UADE or SAE, the |
| | Sponsor Medical Monitor may unmask the treatment regimen |
| | of subject(s) and may discuss this with the Principal |
| | Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | Eye-Cept Rewetting drops, lens cases, glass vials, saline, |
| Specific Materials | ETDRS light cabinet, logMAR charts, and Near logMAR |
| | charts. Optifree®Replenish® Contact Solution. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience

BCC Binocular Crossed Cylinder BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CLDEQ-8 Contact Lens Dry Eye Questionnaire-8

CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Council for Harmonization
IDE Investigational Device Exemption

IEC Independent Ethics Committee
IRB Institutional Review Board

IRB Institutional Review Board

ISO International Organization for S

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution

LSM Least Square Means

MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eve

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye OU Both Eyes PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision recently launched a multifocal contact lens, 1-DAY ACUVUE® Moist Multifocal. The lens is the only marketed soft multifocal lens to have its optical design optimized for the changes that occur in pupil size with refractive error. The modality for the lens is daily disposable. There is a desire to evaluate the same optical design in a reusable modality. The purpose of this study is to evaluate a multifocal optical design manufactured from senofilcon-A material and compare the visual performance to the 1-DAY ACUVUE® Moist Multifocal.

# 1.1. Name and Descriptions of Investigational Products

Test Lens: JJV Investigational senofilcon-A Multifocal Contact Lens-The lens has the same optical design, diameter, base curve and aspheric back surface design as the 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal. The lens is manufactured in senofilcon-A.

Control Lens: Marketed 1-Day Acuvue® Moist Brand Multifocal Contact Lenses

# 1.2. Intended Use of Investigational Products

Both lenses are intended to correct spherical refractive error and presbyopia. The Test lenses are intended to be used as a 2-week, reusable, daily wear lens. The lenses require use of a care system to clean and disinfect the lenses. The control lenses are daily wear lenses that are disposed of at the end of each wear cycle. No care system is required for the control lenses.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding JJV investigational senofilcon-A multifocal refer to the latest version of the Investigator Brochure.

# 1.4. Summary of Known Risks and Benefits to Human Subjects

The Investigational multifocal contact lenses are designed as a continuous asphere providing for the correction of refractive spherical ammetropia and presbyopia. The material is a silicone hydrogel material, senofilcon-A.

The 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens is a currently marketed product that is made of the etafilcon-A material. The contact lenses are available as continuous aspheres providing for the correction of a subjects refractive spherical ammetropia and presbyopia.

The intent of the Test lens is daily wear, reusable lens that the subject wears while awake. This lens is not intended for extended wear. Anticipated risks and adverse reactions with this lens are similar to other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the Section 13 of this protocol. The investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. For the most comprehensive clinical information regarding the JJV

Investigational senofilcon-A multifocal lens refer to the Investigator Brochure. Additional details on the 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens can be found in the package insert in Appendix C.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

The study was a dispensing clinical trial with primary end points of logMAR visual acuity at fit and CLUE vision scores at 1 week. The study was a cross-over design with a marketed product serving as the control. Subjects were fit in the lenses and wore them for 2-4 then attended the first follow-up visit to determine if lens optimization was required. The lenses were than worn for an additional 2 weeks with a 1-week follow-up during that period. There were 32 subjects that completed the study as cohort. The Test lens displayed good visual acuity with the mean distance and intermediate logMAR acuity better than 0.0 and the mean near logMAR acuity better than +0.1 logMAR. This with true of the acuity at the initial fit as well as the 1 week and 2-week visits in the final lens pair. There were two non-ocular adverse events that occurred during the study that were not related to any of the Test lenses.

which at the writing of this protocol has completed data collection, however does not have a completed clinical study report. During the study there were no serious adverse events reported.

In addition to the above study, JJV had tested similar optical designs that have been manufactured in a similar material however those lenses were worn as daily disposable lenses.

was a non-dispensing evaluation with a primary endpoint of logMAR visual acuity. There were 22 subjects that completed the trial per protocol. In this study, the lenses provided clinically acceptable visual acuity with the mean bright high contrast binocular logMAR acuity of -0.016, -0.028 and 0.086 for distance, intermediate and near respectively. There were no adverse events reported during the study.

was a dispensing clinical trial with the primary endpoint of logMAR visual acuity. There were 21 subjects that completed the trial per protocol. The lenses displayed clinically acceptable logMAR visual acuity after approximately 10 days of wear with the mean bright high contrast binocular logMAR acuity of -0.082, -0.042 and 0.054 for distance, intermediate and near respectively. There were two adverse events reported during the study one that was non-ocular and not related to the test articles the other was an ocular adverse event, contact lens induced peripheral ulcer, that was classified as likely related to the study lens. The event resolved with treatment and the subject was discontinued from the study. For additional details refer to the Investigator Brochure for this study.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

# 2.1. Objectives

This study is an evaluation of the visual performance, subjective response, lens fit and ocular physiological response of the JJV Investigational senofilcon A Multifocal Contact Lens. The Test lenses will be compared to the 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens manufactured in etafilcon A material for CLUE subjective vision.

# Primary Objective

This study is an evaluation of how the subjective response of the JJV Investigational senofilcon A Multifocal Contact Lens compares to the 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens manufactured in etafilcon A material.

# 2.2. Endpoints

The study endpoints will be the subjective CLUE Vision scores. Additional endpoints will be logMAR visual acuity at distance, intermediate and near a summary of lenses needed to fit (optimize) the subject, CLUE comfort/handling scores, the lens fit and ocular physiological responses.

#### **Primary Endpoints**

• CLUE vision scores

#### Other Observation(s)

- LogMAR visual acuity scores
- Lens fit
- Corneal staining
- Ocular redness (bulbar and limbal)
- Summary of lenses needed to fit (optimize) the subject
- CLUE comfort/handling scores
- PRO individual questions

#### 2.3. Hypotheses

The following primary hypothesis will be tested throughout this investigation.

#### **Primary Hypothesis:**

1. After 14 to 20 days of wear, the PRO CLUE vision score for the Test lenses will be statistically better than 32 points. This will be recorded by the subject using the CLUE Follow-up Questionnaire.

If the primary hypothesis is met, the following secondary hypothesis will be tested.

# Secondary Hypothesis:

1. After 14 to 20 days of wear, the PRO CLUE vision score for the Test lenses will be non-inferior to the control lens. A non-inferiority margin of 5 CLUE points will be used. This will be recorded by the subject using the CLUE Follow-up Questionnaire.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. They will be hyperopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be between 40 and 70 years of age (inclusive).
- 4. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 5. The subject's refractive cylinder must be  $\leq$ 0.75 D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 7. The subject must have distance best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.
- 8. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
- 10. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea,

- Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 7. A history of amblyopia, strabismus or binocular vision abnormality.
- 8. Any current ocular infection or inflammation.
- 9. Any current ocular abnormality that may interfere with contact lens wear.
- 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.
- 11. Use of any ocular medication, with the exception of rewetting drops.
- 12. History of herpetic keratitis.
- 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 15. Any known hypersensitivity or allergic reaction to Optifree<sup>®</sup>Replenish<sup>®</sup> multipurpose care solution or Eye-Cept<sup>®</sup> rewetting drop solution.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The clinical study is a randomized-controlled, single-masked, cross-over clinical trial. There are two study treatments. A total of approximately 60 eligible hyperopic subjects will be targeted to complete the study. Each Test article will be dispensed for  $3\pm1$  days and an optimization visit will occur. The final lens pair will be dispensed for  $7\pm1$  days and the first follow-up on the final lens pair will occur. The lenses will be dispensed for an additional  $7\pm1$  days and the final lens measurements will be made. The second study lenses will then be fit and the above sequence repeated.

# 4.2. Study Design Rationale

The study is intended to compare two study lens types and the initial performance, in terms of the subjective response after a period of lens dispensing. The lenses are dispensed to determine the subjective responses and the comparison is made after a total of 14-20 days of wear.

The cross-over study design was chosen to control for variables that may impact the lens performance between subjects. It was determined that a washout was not required as previous studies on similar populations with similar multifocal designs did not show a significant carry over effect on the primary/secondary endpoints measured in the study.

#### 4.3. Enrollment Target and Study Duration

A total of approximately 70 eligible subjects will be enrolled with 60 targeted to complete the study.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design with 2 lens types and 2 periods. Using a computer-generated randomization scheme provided by the study biostatistician, each subject will randomly be assigned to one of two unique sequences (Test/Control or Control/Test). Randomization will be stratified by site.

Permuted block randomization will be used to avoid bias in the assignment of subjects to treatment, and to enhance the validity of statistical comparisons across treatment groups. Each block will contain two different lens trial sequences.

The order of lens wear will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

#### 5.2. Masking

This is a single-masked study with the subjects being masked. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

# 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test | | Control | |
|---|---|---|---|---|
| Name | JJV Investigational<br>Multifocal Contact<br>Lens | ACUVUE OASYS® 2-WEEK with HYDRACLEAR® PLUS | 1-Day Acuvue®<br>Moist Brand<br>Multifocal Contact<br>Lens | 1-Day Acuvue <sup>®</sup><br>Moist Brand<br>Contact Lens |
| Manufacturer | Johnson & Johnson®<br>Vision, Inc. | Johnson &<br>Johnson® Vision,<br>Inc. | Johnson &<br>Johnson® Vision,<br>Inc. | Johnson &<br>Johnson® Vision,<br>Inc. |
| | | Over labeled | Over labeled | Over labeled |
| Lens Material | senofilcon A | senofilcon A | etafilcon A | etafilcon A |
| Nominal Base<br>Curve @ 22 °C | 8.35 mm | 8.4 | 8.4 mm | 8.5 |
| Nominal<br>Diameter @ 22 °<br>C | 14.3 mm | 14.0 | 14.3mm | 14.2 |
| Nominal<br>Distance Powers<br>(D) | +1.00 D to<br>+4.00 D in 0.25 D<br>steps | +1.00 D to<br>+4.00 D in 0.25 D<br>steps | +1.00 D to +4.00 D<br>in 0.25 D steps | +1.00 D to +4.00 D<br>in 0.25 D steps |

| | Test | | Control | |
|---|---|---|---|---|
| Nominal | None | None | None | None |
| Cylinder Powers | | | | |
| (D) and Axes | | | | |
| Nominal ADD | Low, Mid, High | None | Low, Mid, High | None |
| Powers (D) | | | | |
| Water Content | 38% | 38% | 58% | 58% |
| Center Thickness | $0.070~\mathrm{mm}$ | 0.070 mm | 0.084 mm | 0.084 mm |
| | (-3.00 D) | (-3.00 D) | (-3.00 D) | (-3.00 D) |
| Oxygen | 122.0 | 122.0 | 28.0 | 28.0 |
| Permeability | | | | |
| (Dk) | | | | |
| Wear Schedule | Daily Wear | Daily Wear | Daily Wear | Daily Wear |
| in Current Study | Reusable | Reusable | | |
| Replacement | Two Weeks | Two Weeks | Daily Disposable | Daily Disposable |
| Frequency | | | | |
| Packaging Form | Blister | Blister | Blister | Blister |
| (vial, blister, | | | | |
| etc.) | | | | |

# 6.2 Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution | |
|---|---|---|
| Solution<br>Name/Description | Eye-Cept® Rewetting<br>Drops | OPTI-FREE® Replenish®<br>Multipurpose Disinfecting<br>Solution |
| Manufacturer | Optics Laboratory | Alcon Laboratories |
| Preservative | Non-Preserved | Myristamidopropyl<br>dimethylamine 0.0005%<br>polyquaternium-1 0.001% |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



# **6.5.** Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

# 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJV.

#### 6.7. Accountability of Test Articles

JJV will provide the Investigator with sufficient quantities of study article and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to the Sponsor.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

Site Instructions for Test Article Receipt and Test Article Accountability for additional information

# 7. STUDY EVALUATIONS

# 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment 1 | Treatment 2 | Treatment 2 | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Follow-up 3 | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| | Treatment 1 | Optimization | | Treatment 2 | Optimization | | |
| | | | | Fitting | | | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 | from V6 |
| | | | | Fitting Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours | 1.5 hours |
| Duration | | | | | | | |
| Statement of | | | | | | | |
| Informed Consent | X | | | | | | |
| Demographics | X | | | | | | |
| Medical | | | | | | | |
| History/Concomitant | | | | | | | |
| Medications | X | | | | | | |
| Adverse Events and | | | | | | | |
| Concomitant | | | | | | | |
| Medications Review | | X | x | X | X | X | X |
| Compliance | | X | X | X | X | X | X |
| Habitual Contact | | | | | | | |
| Lens Information | X | | | | | | |
| Contact Lens | | | | | | | |
| History | X | | | | | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment 1 | Treatment 2 | Treatment 2 | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Follow-up 3 | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| | Treatment 1 | Optimization | | Treatment 2 | Optimization | | |
| | | | | Fitting | | | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 | from V6 |
| | | | | Fitting Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours | 1.5 hours |
| Duration | | | | | | | |
| Wear Time and | | | | | | | |
| Comfortable Wear | | | | | | | |
| Time with lenses | X | X | X | X | X | X | X |
| Screening | | | | | | | |
| Inclusion/Exclusion | | | | | | | |
| Criteria | X | | | | | | |
| Subject Reported | | | | | | | |
| Ocular Symptoms | X | X | X | X | X | X | X |
| Baseline | | | | | | | |
| Questionnaire | X | | | | | | |
| CLDEQ-8 | | | | | | | |
| Questionnaire | X | | X | X | | X | X |
| Distance and Near | | | | | | | |
| Entrance Visual | | | | | | | |
| Acuity | X | X | X | X | X | X | X |
| Lens Removal | X | X | X | X | X | X | X |
| Keratometry | X | | | | | | |
| Subjective | | | | | | | |
| Refraction and | | | | | | | |
| Distance Visual | | | | | | | |
| Acuity | X | | | | | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment 1 | Treatment 2 | Treatment 2 | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Follow-up 3 | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| | Treatment 1 | Optimization | • | Treatment 2 | Optimization | • | • |
| | | 1 | | Fitting | 1 | | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 | from V6 |
| | | | | Fitting Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours | 1.5 hours |
| Duration | | | | | | | |
| Near ADD | | | | | | | |
| Determination | X | | | | | | |
| Ocular Dominance | X | | | | | | |
| ADD Refinement | X | | | | | | |
| Near Visual Acuity | X | | | | | | |
| Biomicroscopy | X | X | X | X | X | X | X |
| Baseline | | | | | | | |
| Inclusion/Exclusion | | | | | | | |
| Criteria | X | | | | | | |
| Continuance | | | | X | | | |
| Lens Selection | X | | | X | | | |
| Lens Insertion | X | X | X | X | X | X | |
| 10 Minute Settling | X | X | | X | X | | |
| Visual Satisfaction / | | | | | | | |
| Subjective | | | | | | | |
| Acceptance | X | X | X | X | X | X | X |
| Study Lens Distance | | | | | | | |
| and Near Visual | | | | | | | |
| Acuity | X | X | X | X | X | X | X |
| Distance Over | X | X | | X | X | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment 1 | Treatment 2 | Treatment 2 | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Follow-up 3 | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| | Treatment 1 | Optimization | | Treatment 2 | Optimization | | |
| | | | | Fitting | | | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 | from V6 |
| | | | | Fitting Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours | 1.5 hours |
| Duration | | | | | | | |
| Refraction and | | | | | | | |
| Visual Acuity | | | | | | | |
| Subjective Lens Fit | | | | | | | |
| Assessment | X | X | X | X | X | X | X |
| Binocular Over | | | | | | | |
| Refraction | | | X | X | | X | X |
| Visual Performance | | | X | X | | X | X |
| Modifications | X | X | | X | X | | |
| Post-Fit | | | | | | | |
| Questionnaire | X | X | | X | X | | |
| Worn Lens | | | | | | | |
| Collection | | X | | X | X | | X |
| PRO Questionnaire | X | X | X | X | X | X | X |
| Distance and Near | | | | | | | |
| Exit Visual Acuity | X | X | X | X | X | X | X |
| Dispensing Criteria | X | X | X | X | X | X | |
| Instructions | X | X | X | X | Х | X | |
| Schedule Follow-up | X | X | X | X | X | X | |
| Final Evaluation | | | | | | | X |

# 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline CLUE performance. If the subject is not wearing their lenses they must be rescheduled.

| | | Visit 1: Screening |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.6 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subjects wear time and comfortable wear time with their habitual contact lenses. |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.8 | Baseline and<br>CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO questions. |

| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended | |
|---|---|---|---|
| 1.10 | T ( TT 1 | symptoms questionnaire. | |
| 1.10 | Entrance Visual | Distance and near Snellen visual acuity will be | |
| | Acuity | measured for each eye with the subject's | |
| | | habitual contact lenses in place. | |
| | | For near measures use the ETDRS 2000 Series | |
| | | Chart 1 or 2. The acuity will be recorded to | |
| | | the nearest letter OD, OS and OU. | |
| 1.11 | Lens Removal | Have the subject remove their habitual lenses | |
| | | and store in an approved storage solution. | |
| 1.12 | Keratometry | Keratometry will be performed OD and OS | |
| | | and the steep and flat dioptric power and | |
| | | corresponding meridians recorded. | |
| 1.13 | Subjective Refraction | An optimal, binocular balanced distance | |
| | and Distance Visual | sphero-cylindrical refraction will be | |
| | Acuity | performed. Record the refraction and distance | |
| | | visual acuity to the nearest letter. | |
| | | Note: Best distance visual acuity with sphero- | |
| | | cylindrical refraction must be at least 20/20 <sup>-3</sup> | |
| | | in each eye for the subject to be eligible in the | |
| | | study. | _ |
| 1.14 | Near ADD | The near reading addition will be determined | |
| | Determination | using the binocular crossed cylinder technique | |
| | | (BCC) at 40 cm followed by optimization in a | |
| 1.15 | Ocular Dominance | trial frame in step 1.16 below. Determine the distance ocular dominance with | Annandiy E |
| 1.13 | Ocular Dominance | | Appendix F |
| | | the best distance correction in place using a +1.00-blur test. If the results are equivocal use | |
| | | the sighting dominance test to determine the | |
| | | dominant eye used for the study. | |
| 1.16 | ADD Refinement | Place the BCC result in the trial frame and | |
| | | refine the near prescription with trial lenses (or | |
| | | flippers) under binocular conditions. | |
| 1.17 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 | |
| | | near card placed at 40 cm. Record the near | |
| | | visual acuity OD, OS and OU at 40 cm. | _ |
| 1.18 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine | |
| | | eligibility. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | 1 | be graded in 1.0 increments. | |

| | | If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
|---|---|---|
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 1.19 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If so, proceed to lens fitting. If not, complete the final evaluation and discharge the subject. |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.20 | Randomization and | Record the randomization ID and lens wear | |
| | Lens Wear Schedule | schedule (daily disposable, daily reusable | |
| 1.01 | T 0.1 / | wear). | Α 1' |
| 1.21 | Lens Selection | Select the lens pair and power based on the | Appendix<br>G and H |
| | | Randomization and fitting guide for each eye. | (Fitting |
| | | Record the test lens parameters (power and lot number). | Guides) |
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If | Guides) |
| 1.22 | Lens insertion | the lens is uncomfortable, inspect for damage | |
| | | and remove, reinsert or replace as necessary. | |
| | | Damaged lenses will be stored in labeled vial | |
| | | with sterile saline, and clearly differentiated | |
| | | from the other worn lenses that will be shipped | |
| | | back to the Sponsor. Complete the Quality | |
| | | Product Complaint form. | |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum | |
| | | of 10 minutes. | |
| 1.24 | Determine Visual | Determine if the subject's vision is acceptable | |
| | Satisfaction | with the lenses. Allow the subject to look | |
| | | down a hallway or out of a window for | |
| | | distance vision assessments, and for them to | |
| | | read a book, magazine or similar for near vision. | |
| 1.25 | Study Lens Distance | Measure the distance and near visual acuity | |
| 1.23 | and Near Visual | OD, OS and OU. Record the results. | |
| | Acuity | ob, ob and ob. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or | |

| | | 2 near card placed at 40 cm to measure the | |
|---|---|---|---|
| | | Near visual acuity | |
| 1.26 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.27 | Subjective Lens Fit<br>Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> | |
| 1.28 | Modifications | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. | Appendix G and H (Fitting Guides) |

| | 1 | T |
|---|---|---|
| | | If modifications are required steps 1.21-1.27 will be repeated for each modification. |
| 1.29 | Post-Fit | The subject will evaluate the vision |
| 1.27 | Questionnaire | characteristics, comfort characteristics, |
| | Questionnaire | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| | | questionnaire. |
| 1.30 | Distance and Near | Distance and near Snellen visual acuity will be |
| 1.50 | Exit Visual Acuity | measured for each eye with the study contact |
| | | lenses in place. |
| | | For near measures use the ETDRS 2000 Series |
| | | Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| | | · |
| | | Note: The distance visual acuity must be at |
| | | least 20/30 OU for the lenses to be |
| | | dispensed. |
| 1.31 | Dispensing Criteria | The lenses will be dispensed for 2-4 days. |
| | | Distance Snellen acuity equal to or better |
| | | than 20/30 OU |
| | | • Subject must indicate that the vision is |
| | | acceptable. |
| | | • Subject must indicate that the comfort of |
| | | the lenses is acceptable. |
| | | Lenses must have an acceptable general |
| | | lens fit. |
| 1.32 | Patient Instructions | Instruct the Subject the following: |
| | for Daily Disposable | The lenses will be worn on a daily wear |
| | Lenses | basis. |
| | | Only enough lenses will be dispensed to |
| | | the subject to wear for the required number |
| | | of days until their follow-up visit. No |
| | | additional lenses will be dispensed. |
| | | A new lens will be opened and worn each |
| | | day. |
| | | • Instruct the subject to bring back all |
| | | unworn study lenses. |
| | | No cleaning or disinfecting solutions will |
| | | be used. If determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |
| | | ased as needed for dryness. |

# • Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.

- Subjects will be instructed to wear their glasses when not wearing the study lenses.
- A patient instruction booklet will be provided.

Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.

# 1.33 Patient Instructions for Daily Reusable Wear Lenses

Instruct the Subject the following:

- The lenses will be worn on a daily wear basis.
- OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.
- If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.
- Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.
- Subjects will be instructed to wear their glasses when not wearing the study lenses.
- A patient instruction booklet will be provided.

Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint

| | | Form. The lens will be stored in labeled vial |
|---|---|---|
| | | with sterile saline, and returned to the |
| | | Sponsor. |
| 1.34 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 day. |
| | | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

# VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 2: Treatment 1 Follow-up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history |
| 2.2 | Wear Time | changes from the previous study visit. Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 2.4 | PRO Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 2.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.6 | Subjective<br>Acceptance | Record whether the subjects distance and near vision with the lenses is acceptable. |
| 2.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Note: Use the ETDRS 2000 Series Chart 1 or |

| | T | T | |
|---|---|---|---|
| | | 2 near card placed at 40 cm to measure the | |
| 2.0 | D' . O | Near visual acuity | |
| 2.8 | Distance Over- | Perform a distance over-refraction OD and OS | |
| | Refraction and | using loose lenses outside of the phoropter | |
| | Distance Visual | under ambient room illumination. The | |
| | Acuity | distance over-refraction may also be refined | |
| | | under binocular conditions. Record the results | |
| | | and distance visual acuity OD and OS. | |
| | | The results of the distance over-refraction may | |
| | | also be checked for the impact on near vision | |
| 2.0 | D | under monocular and/or binocular conditions. | A 1. |
| 2.9 | Determination of | If the subject reports unsatisfactory vision, or is | Appendix |
| | Lens Optimization | unable to obtain 20/30 distance visual acuity<br>OU with the lenses then a modification must be | G and H |
| | | | (Fitting |
| | | attempted. If the subject reports satisfactory vision with | Guides) |
| | | If the subject reports satisfactory vision with the lenses a modification is not required, | |
| | | however at the Investigator's discretion and | |
| | | based upon their findings on the measured | |
| | | visual acuity and/or over- refraction the | |
| | | investigator may make a modification. | |
| | | Up to two attempts at modification are | |
| | | permitted if necessary, in order to achieve an | |
| | | acceptable distance and near binocular | |
| | | performance for the subject, and to enable | |
| | | them to wear that particular lens type. | |
| | | Follow the fitting guide allowing for at least | |
| | | 10 minutes of settling time between each lens | |
| | | modification attempted. | |
| 2.10 | Lens Fit Assessment: | Evaluate and grade lens centration, primary | |
| | | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | • The subject should not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | • presence of limbal exposure (appearance of | |
| | | clear cornea) in any gaze | |
| | | • presence of edge lift | |
| | | presence of unacceptable movement | |
| | | (excessive or insufficient) in all three | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |
| | | evaluation, and complete the Final Evaluation | |
|---|---|---|--|
| 2.11 | Collection of unworn lenses (if applicable) | form. Collect unworn lenses returned by the subject when lens power has been optimized | |
| | renses (ir applicable) | Note: If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 1 and dispense enough lenses of the same | |
| | | power to last the subject until their next visit. | |
| 2.12 | Lens Removal | The study lenses will be removed and discarded. | |
| 2.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness unit increments will be used in the grading. | |
| | | Corneal Staining Assessment (CTP-2003) will be graded in 1.0 increments. If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops or saline may be instilled. | |
| 2.14 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 2.12 above. | |
| 2.15 | PRO Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. | |
| 2.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| | | Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. | |
| 2.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 7±1 day.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is</li> </ul> | |
| | | acceptable. | |

| 2.18 | Patient Instructions for Daily Disposable Lenses | <ul> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved</li> </ul> |
|---|---|---|
| | | <ul> <li>rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.</li> </ul> |
| 2.19 | Patient Instructions<br>for Daily Reusable<br>Wear Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Replenish® solution will be</li> </ul> |

| 2.20 | Schedule | used in a rub regime to disinfect and store the lenses each night in the lens case provided. • If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. • Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. • Subjects will be instructed to wear their glasses when not wearing the study lenses. Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. The subject will be scheduled to return for |
|---|---|---|
| 2.20 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and | Review the subject's concomitant medications |
| | Concomitant | and record any changes from the previous |
| | Medications Review | study visit. |
| | | Record any adverse events or medical history |
| | | changes from the previous study visit. |
| 3.2 | Wear Time | Record the hours the subject has worn the |

| | | study lenses and the comfortable wear time on |
|---|---|---|
| | | the day of follow-up. |
| 3.3 | Compliance | Record the subject's compliance with wearing the study lenses. |
| | | Note: Subjects must have worn lenses for at least 6 hours per day |
| | | To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 |
| | | hours prior to the visit. |
| 3.4 | PRO and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 3.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 3.6 | Subjective | Record whether the subjects distance and near |
| | Acceptance | vision with the lenses is acceptable. |
| 3.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. |
| | 1200219 | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 3.8 | Visual Performance<br>Distance (3M) | Visual performance will be recorded <b>OU</b> for the following: |
| | Intermediate (64 cm) | Distance, Bright Illuminance |
| | Near (40 cm) | ETDRS Charts 3M-HC#3 and LC#3 |
| | | Near, Bright Illuminance |
| | | Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast (1 Chart) and Low Contrast (1 Chart). |
| | | Near (40 cm) High Contrast (1 Chart) and Low Contrast (1 Chart). |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) |
| | | ETDRS Charts 3M-HC#6 |
| | | Near, Dim Illuminance (with <u>Near</u> goggles) |
| | | Reduced Guillon-Poling charts |
| | | High Contrast (1 Chart at each distance)<br>Intermediate (64 cm) and Near (40 cm). |
| | | Note: |

| | | <ul> <li>The room illuminance must be between 7.3 and 7.9 EV.</li> <li>Distance, HC-1 Chart luminance Acceptable EV Range 10.5-10.7.</li> <li>Guillon-Poling, Near Chart Luminance Acceptable EV Range 10.8-11.1.</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be</li> </ul> | |
|---|---|---|---|
| 3.9 | Binocular Distance | simulated by using the goggles) Perform a binocular over-refraction and record | Appendix |
| | Over-refraction and<br>Distance Visual<br>Acuity | the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | D D |
| 3.10 | Lens Fit Assessment: | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> | |
| 3.11 | Lens Removal | Have the subject wearing the daily disposable lenses remove and discard the lenses. Subjects that are wearing the daily wear lens will remove and temporarily store in a lens case in OPTI-FREE® Replenish® to be reinserted after biomicroscopy. | |
| 3.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp<br>Classification Scales will be used to grade the<br>findings.<br>For the conjunctival redness 0.5 | |

| | | unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
|---|---|---|
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 3.13 | Insertion of Study<br>Lenses | Dispense the subject new lenses if wearing the daily disposable lenses that match the Distance and ADD power of the lenses that were removed in Step 3.11 above. |
| | | Subjects that are wearing the daily reusable wear lenses will reinsert the lenses that were temporarily stored. |
| 3.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at |
| | | least 20/30 OU for the lenses to be dispensed. |
| 3.15 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 7±1 day.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 3.16 | Patient Instructions for Daily Disposable Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> </ul> |

# Instruct the subject to bring back all unworn study lenses. No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. • Subjects will be instructed to wear their glasses when not wearing the study lenses. *Note:* In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. 3.17 **Patient Instructions** Instruct the Subject the following: for **Daily Reusable** The lenses will be worn on a daily wear **Wear Lenses** • OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided. • If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. Subjects will be instructed to wear their glasses when not wearing the study lenses. *Note:* In the event a lens is lost or damaged, the subject will return to the investigator site

| | | for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
|---|---|---|
| 3.18 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 4 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 4: Treatment 1 Follow-up 3 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and | Review the subject's concomitant medications |
| | Concomitant | and record any changes from the previous |
| | Medications Review | study visit. |
| | | Record any adverse events or medical history |
| | | changes from the previous study visit. |
| 4.2 | Wear Time | Record the hours the subject has worn the |
| | | study lenses and the comfortable wear time on |
| | | the day of follow-up. |
| 4.3 | Compliance | Record the subject's compliance with wearing |
| | | the study lenses. |
| | | Note: Subjects must have worn lenses for at |
| | | least 6 hours per day |
| | | To be counted as a day of wear at this visit the |
| | | Subject must have worn the study lenses for 6 |
| | | hours prior to the visit. |
| 4.4 | PRO and CLDEQ-8 | The subject will evaluate the vision |
| | Questionnaires | characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| | | questionnaire. |
| 4.5 | Subject Reported | Subjects will respond to a verbal open-ended |
| | Ocular Symptoms | symptoms questionnaire. |
| 4.6 | Distance and Near | Distance and near Snellen visual acuity will be |
| | Entrance Visual | measured for each eye with the study contact |

| | Acuity | lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
|---|---|---|---|
| 4.7 | Visual Performance<br>Distance (3M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance ETDRS Charts 3M-HC#1, HC#2, HC#3 and LC#1, LC#2 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts High Contrast and Low Contrast Intermediate (64 cm) and | |
| | | Near (40 cm). Distance, Dim Illuminance (with <u>Distance</u> goggles) | |
| | | ETDRS Charts 3M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with Near goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). | |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV.</li> <li>Distance, HC-1 Chart luminance Acceptable EV Range 10.5-10.7.</li> <li>Guillon-Poling, Near Chart Luminance Acceptable EV Range 10.8-11.1.</li> <li>Do not use the Mesopic filter for Dim</li> </ul> | |
| 4.8 | Binocular Distance<br>Over-refraction and<br>Distance Visual | luminance (Dim luminance will be simulated by using the goggles). Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed | Appendix<br>D |
| 4.9 | Acuity Lens Fit Assessment: | based on the over-refraction. Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze | |

| | | • |
|---|---|---|
| | | presence of edge lift |
| | | presence of unacceptable movement |
| | | (excessive or insufficient) in all three |
| | | movement categories (primary gaze, |
| | | upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the |
| | | subject will be discontinued from the study. |
| | | Remove the lenses, perform a slit-lamp |
| | | evaluation, and complete the Final Evaluation |
| | | form. |
| 4.10 | Lens Removal | Have the subject remove the study lenses and |
| | | store in saline in a labeled glass vial. |
| | | Note: Lenses do not need to be stored in a |
| | | refrigerator. |
| 4.11 | Biomicroscopy | FDA Slit Lamp Classification Scale will be |
| | | used to grade the findings and determine |
| | | eligibility. |
| | | For the conjunctival redness 0.5 |
| | | unit increments will be used in the grading. |
| | | Corneal Staining Assessment will will |
| | | be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be |
| | | expedited, preservative-free rewetting drops or |
| 1.10 | | saline may be instilled. |
| 4.12 | Continuance | Determine whether the subject is eligible to |
| | | continue in the study based on the examination findings. |
| | | mungs. |

| | Visit 4: Treatment 2 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.13 | Lens Wear Schedule | Record the lens wear schedule (daily disposable, daily reusable wear). | |
| 4.14 | Lens Selection | Select the lens pair and power based on the Randomization and fitting guide for each eye. Record the Test lens parameters (power and lot number). | Appendix G and H (Fitting Guides) |
| 4.15 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated | · |

| | T | | |
|---|---|---|---|
| | | from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. | |
| 4.16 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 4.17 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 4.18 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 4.19 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 4.20 | Subjective Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation | |
| 4.21 | Modifications | form. If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity | Appendix G (Fitting |

| 4.22 | Post-Fit | OU with the lenses then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 4.14-4.20 will be repeated for each modification The subject will evaluate the vision | Guide) |
|---|---|---|---|
| | Questionnaire | characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. | |
| 4.23 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. | |
| 4.24 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 2-4 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> | |
| 4.25 | Patient Instructions<br>for <b>Daily Disposable</b><br><b>Lenses</b> | <ul><li>Instruct the Subject the following:</li><li>The lenses will be worn on a daily wear basis.</li></ul> | |

# Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. A new lens will be opened and worn each Instruct the subject to bring back all

- unworn study lenses.
- No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.
- Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.
- Subjects will be instructed to wear their glasses when not wearing the study lenses.
- A patient instruction booklet will be provided.

*Note:* In the event a lens is lost or damaged. the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.

#### 4.26 **Patient Instructions** for Daily Reusable **Wear Lenses**

Instruct the Subject the following:

- The lenses will be worn on a daily wear basis.
- OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.
- If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.
- Subjects will be instructed to wear lenses

| | | for a minimum of 6 hours a day, every day |
|---|---|---|
| | | during the study. |
| | | Subjects will be instructed to wear their glasses when not wearing the study lenses. |
| | | A patient instruction booklet will be provided. |
| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile |
| | | saline, and returned to the Sponsor. |
| 4.27 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 day. |
| | | Note: To count the follow-up visit as a day of wear the Subject must have worn the study |
| | | lenses for 6 hours prior to the visit. |

The subjects must present to Visit 5 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | | Visit 5: Treatment 2 Follow-up 1 |
|---|---|---|
| Step | Procedure | Details |
| 5.1 | Adverse Events and | Review the subject's concomitant medications |
| | Concomitant | and record any changes from the previous |
| | Medications Review | study visit. |
| | | Record any adverse events or medical history |
| | | changes from the previous study visit. |
| 5.2 | Wear Time | Record the hours the subject has worn the |
| | | study lenses and the comfortable wear time on |
| | | the day of follow-up. |
| 5.3 | Compliance | Record the subject's compliance with wearing |
| | | the study lenses. |
| | | Note: Subjects must have worn lenses for at |
| | | least 6 hours per day |
| | | To be counted as a day of wear at this visit the |
| | | Subject must have worn the study lenses for 6 |
| | | hours prior to the visit. |
| 5.4 | PRO Questionnaire | The subject will evaluate the vision |

| | | characteristics, comfort characteristics, | |
|---|---|---|---|
| | | handling characteristics, and visual symptoms | |
| | | of the study lenses using the PRO | |
| 5.5 | Ogular Symptoma | questionnaire. | |
| 3.3 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire | |
| 5.6 | Subjective | Record whether the subjects distance and near | |
| | Acceptance | vision with the lenses is acceptable. | |
| 5.7 | Distance and Near | Distance and near Snellen visual acuity will be | |
| | Entrance Visual | measured for each eye with the study contact | |
| | Acuity | lenses in place. | |
| | | For near measures use the ETDRS 2000 Series | |
| | | Chart 1 or 2. The acuity will be recorded to the | |
| | | nearest letter OD, OS and OU. | |
| 5.8 | Distance Over- | Perform a distance over-refraction OD and OS | |
| | Refraction and | using loose lenses outside of the phoropter | |
| | Distance Visual | under ambient room illumination. The | |
| | Acuity | distance over-refraction may also be refined | |
| | | under binocular conditions. Record the results | |
| | | and distance visual acuity OD and OS. The | |
| | | results of the distance over-refraction may also | |
| | | be checked for the impact on near vision under | |
| 5.9 | Determination of | monocular and/or binocular conditions. If the subject reports unsatisfactory vision, or is | Ammondia |
| 3.9 | | unable to obtain 20/30 distance visual acuity | Appendix G and H |
| | Lens Optimization | OU with the lenses then a modification must be | (Fitting |
| | | attempted. | Guides) |
| | | If the subject reports satisfactory vision with | Guides) |
| | | the lenses a modification is not required, | |
| | | however at the Investigator's discretion and | |
| | | based upon their findings on the measured | |
| | | visual acuity and/or over- refraction the | |
| | | investigator may make a modification. | |
| | | Up to two attempts at modification are | |
| | | permitted if necessary, in order to achieve an | |
| | | acceptable distance and near binocular | |
| | | performance for the subject, and to enable | |
| | | them to wear that particular lens type. | |
| | | Follow the fitting guide allowing for at least 10 minutes of settling time between each lens | |
| | | modification attempted. | |
| 5.10 | Lens Fit Assessment: | Evaluate and grade lens centration, primary | |
| | | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | The subject should not proceed to wear the | |

| | | lenses if any of the following is observed: |
|---|---|---|
| | | • presence of limbal exposure (appearance of |
| | | clear cornea) in any gaze |
| | | presence of edge lift |
| | | presence of unacceptable movement |
| | | (excessive or insufficient) in <u>all three</u> |
| | | movement categories (primary gaze, |
| | | upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the |
| | | subject will be discontinued from the study. |
| | | Remove the lenses, perform a slit-lamp |
| | | evaluation, and complete the Final Evaluation |
| | | form. |
| 5.11 | Collection of unworn | Collect unworn lenses returned by the subject |
| | lenses (if applicable) | when lens power has been optimized |
| | | Note: If lens power was not changed allow the |
| | | subject to use the unworn lenses dispensed at |
| | | Visit 4 and dispense enough lenses of the same |
| 5.10 | T D 1 | power to last the subject until their next visit. |
| 5.12 | Lens Removal | The study lenses will be removed and |
| | | discarded. |
| 5.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp |
| | | Classification Scales will be used to grade the |
| | | findings. |
| | | For the conjunctival redness 0.5 |
| | | unit increments will be used in the grading. |
| | | Corneal Staining Assessment will |
| | | be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be |
| | | expedited, preservative-free rewetting drops or |
| | | saline may be instilled. |
| 5.14 | Insertion of Study | Dispense the subject new lenses that match the |
| | Lenses | distance and ADD power of the lenses that |
| | | were removed in Step 5.12 above. |
| 5.15 | PRO Questionnaire | The subject will evaluate the vision |
| | | characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| 5.16 | Distance and Near | questionnaire. |
| 3.16 | | Distance and near Snellen visual acuity will be |
| | Exit Visual Acuity | measured for each eye with the study contact lenses in place. |
| | l | icuses in place. |

| | | For near measures use the ETDRS 2000 Series |
|---|---|---|
| | | Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| | | Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 5.17 | Dispensing Criteria | The lenses will be dispensed for 7±1 day. |
| | Biopensing criteria | <ul> <li>Distance Snellen acuity equal to or better<br/>than 20/30 OU</li> </ul> |
| | | Subject must indicate that the vision is acceptable. |
| | | • Subject must indicate that the comfort of the lenses is acceptable. |
| | | Lenses must have an acceptable general lens fit. |
| 5.18 | Patient Instructions | Instruct the Subject the following: |
| | for Daily Disposable<br>Lenses | The lenses will be worn on a daily wear basis. |
| | | <ul> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> </ul> |
| | | <ul> <li>Instruct the subject to bring back all<br/>unworn study lenses.</li> </ul> |
| | | No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. |
| | | • Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. |
| | | • Subjects will be instructed to wear their glasses when not wearing the study lenses. |
| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably |

| | | possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
|---|---|---|
| 5.19 | Patient Instructions for Daily Reusable Wear Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the</li> </ul> |
| 5.20 | Schedule<br>Follow-up | Sponsor. The subject will be scheduled to return for their follow-up appointment in 7±1 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 6 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | | Visit 6: Treatment 2 Follow-up 2 |
|---|---|---|
| Step | Procedure | Details |
| 6.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 6.2 | Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 6.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 6.4 | PRO Questionnaires<br>and CLDEQ-8 | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 6.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 6.6 | Subjective<br>Acceptance | Record whether the subjects distance and near vision with the lenses is acceptable. |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 6.8 | Visual Performance<br>Distance (3M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded <b>OU</b> for the following: <b>Distance, Bright Illuminance</b> ETDRS Charts 3M-HC#3 and LC#3 <b>Near, Bright Illuminance</b> Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast (1 Chart) and Low |

| | | Contrast (1 Chart). Near (40 cm) High Contrast (1 Chart) and Low Contrast (1 Chart). Distance, Dim Illuminance (with Distance goggles) ETDRS Charts 3M-HC#6 Near, Dim Illuminance (with Near goggles) Reduced Guillon-Poling charts High Contrast (1 Chart at each distance) Intermediate (64 cm) and Near (40 cm). | |
|---|---|---|---|
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV.</li> <li>Distance, HC-1 Chart luminance Acceptable EV Range 10.5-10.7.</li> <li>Guillon-Poling, Near Chart Luminance Acceptable EV Range 10.8-11.1.</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be</li> </ul> | |
| 6.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>D |
| 6.10 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp | |

| | T | | |
|---|---|---|---|
| | | evaluation, and complete the Final Evaluation form. | |
| 6.11 | Lens Removal | Have the subject wearing the daily disposable | |
| 0.11 | Lens Removar | lenses remove and discard the lenses. | |
| | | Subjects that are wearing the daily reusable | |
| | | wear lens will remove and temporarily store in | |
| | | a lens case in OPTI-FREE® Replenish® to be | |
| | | reinserted after biomicroscopy. | |
| 6.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp | |
| | | Classification Scales will be used to grade the | |
| | | findings. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops or | |
| | | saline may be instilled. | |
| 6.13 | Insertion of Study | Dispense the subject new lenses if wearing the | |
| | Lenses | daily disposable lenses that match the Distance | |
| | | and ADD power of the lenses that were | |
| | | removed in Step 6.11 above. | |
| | | Subjects that are wearing the daily wear lenses | |
| | | will reinsert the lenses that were temporarily | |
| | | stored. | _ |
| 6.14 | Distance and Near | Distance and near Snellen visual acuity will be | |
| | Exit Visual Acuity | measured for each eye with the study contact | |
| | | lenses in place. | |
| | | For near measures use the ETDRS 2000 Series | |
| | | Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| | | hearest letter OD, OS and OO. | |
| | | Note: The distance visual acuity must be at | |
| | | least 20/30 OU for the lenses to be | |
| | | dispensed. | |
| 6.15 | Dispensing Criteria | The lenses will be dispensed for 7±1 day. | |
| | | Distance Snellen acuity equal to or better | |
| | | than 20/30 OU | |
| | | Subject must indicate that the vision is | |
| | | acceptable. | |
| | | Subject must indicate that the comfort of | |
| | | 1 | |
| | | the lenses is acceptable. | |

| | | Lenses must have an acceptable general lens fit. |
|---|---|---|
| 6.16 | Patient Instructions for Daily Disposable Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.</li> </ul> |
| 6.17 | Patient Instructions<br>for Daily Reusable<br>Wear Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> </ul> |

| | | <ul> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> </ul> |
|---|---|---|
| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site |
| | | for replacement. As much as reasonably |
| | | possible, a damaged lens should be returned to the investigational site and then returned to |
| | | the Sponsor. If lens damage is present, |
| | | complete the Product Quality Complaint Form. The lens will be stored in labeled vial |
| | | with sterile saline, and returned to the |
| C 10 | C-11-1- | Sponsor. |
| 6.18 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. |
| | 1 onow-up | then follow up appointment in 7±1 days. |
| | | Note: To count the follow-up visit as a day of |
| | | wear the Subject must have worn the study |
| | | lenses for 6 hours prior to the visit. |

The subjects must present to Visit 7 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 7: Treatment 2 Follow-up 3 | |
|---|---|---|
| Step | Procedure | Details |
| 7.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 7.2 | Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 7.3 | Compliance | Record the subject's compliance with wearing the study lenses. |

| | T | |
|---|---|---|
| | | Note: Subjects must have worn lenses for at |
| | | least 6 hours per day |
| | | To be counted as a day of wear at this visit the |
| | | Subject must have worn the study lenses for 6 |
| | PRO 1 CERTO O | hours prior to the visit. |
| 7.4 | PRO and CLDEQ-8 | The subject will evaluate the vision |
| | Questionnaires | characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| | | questionnaire. |
| 7.5 | Subject Reported | Subjects will respond to a verbal open-ended |
| | Ocular Symptoms | symptoms questionnaire. |
| 7.6 | Distance and Near | Distance and near Snellen visual acuity will be |
| | Entrance Visual | measured for each eye with the study contact |
| | Acuity | lenses in place. |
| | | For near measures use the ETDRS 2000 Series |
| | | Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| 7.7 | Visual Performance | Visual performance will be recorded OD, OS, |
| | Distance (3 M) | and OU for the following: |
| | Intermediate (64 cm) | Distance, Bright Illuminance |
| | Near (40 cm) | ETDRS Charts 3M-HC#1, HC#2, HC#3 and |
| | | LC#1, LC#2 and LC#3 |
| | | Near, Bright Illuminance |
| | | Reduced Guillon-Poling Charts High Contrast |
| | | and Low Contrast Intermediate (64 cm) and |
| | | Near (40 cm). |
| | | , , , |
| | | Distance, Dim Illuminance (with <u>Distance</u> |
| | | goggles) |
| | | ETDRS Charts 3M-HC#4, HC#5, HC#6 |
| | | Near, Dim Illuminance (with <i>Near</i> goggles) |
| | | Reduced Guillon-Poling charts |
| | | High Contrast |
| | | Intermediate (64 cm) and Near (40 cm). |
| | | intermediate (or cit) and real (40 cit). |
| | | Note: |
| | | The room illuminance must be |
| | | between 7.3 and 7.9 EV. |
| | | Distance, HC-1 Chart luminance Acceptable EV Pange 10.5.10.7 |
| | | Acceptable EV Range 10.5-10.7. |
| | | Guillon-Poling, Near Chart Lyminance Acceptable EV Pange |
| | | Luminance Acceptable EV Range |
| | | 10.8-11.1 |

| | | Do not use the Mesopic filter for Dim<br>luminance (Dim luminance will be<br>simulated by using the goggles) | |
|---|---|---|---|
| 7.8 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record<br>the OD and OS results and distance visual<br>acuity. Note: No lens changes are allowed based on<br>the over-refraction. | Appendix<br>D |
| 7.9 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 7.10 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. Note: The lenses do not need to be stored in a refrigerator. | |
| 7.11 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Distance Subjective | An optimal, binocular balanced distance |
| | Sphero-cylindrical | sphero-cylindrical refraction will be |
| | Refraction and | performed. |
| | Distance Exit Visual | |
| | Acuity | Record the refraction and distance visual |
| | - | acuity to the nearest letter. |
| F.2 | Subject Disposition | Indicate if the subject completed the study |
| | | successfully. If subject discontinued from the |
| | | study indicate the reason. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Unscheduled Visit | | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for |
| | | reasons for the unscheduled visit |

| | | Unscheduled Visit |
|---|---|---|
| U.2 | Adverse Events and | Review the subject's concomitant |
| | Concomitant Medications | medications and record any changes from |
| | Review | the previous study visit. |
| U.3 | Subject Reported Ocular | Subjects will respond to a verbal open- |
| | Symptoms | ended symptoms questionnaire. |
| U.4 | Entrance VA | Record the entrance distance and near visual |
| | | acuity (OD, OS and OU) to the nearest |
| | | letter. |
| | | For near measures use the ETDRS 2000 |
| | | Series Chart 1 or 2. The acuity will be |
| | | recorded to the nearest letter OD, OS and |
| TIE | Calinatian Calam | OU. |
| U.5 | Subjective Sphero- | An optimal, binocular balanced distance |
| | cylindrical Refraction | sphero-cylindrical refraction will be performed. |
| | | performed. |
| | | Record the refraction and distance visual |
| | | acuity to the nearest letter. |
| U.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be |
| | Біоннеговеору | used to grade the findings and determine |
| | | eligibility. |
| | | For the conjunctival redness 0.5 |
| | | unit increments will be used in the grading. |
| | | Corneal Staining Assessment |
| | | will be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to |
| | | be expedited, preservative-free rewetting |
| 11.5 | T D: : | drops or saline may be instilled. |
| U.7 | Lens Dispensing | Additional study lenses may be dispensed |
| U.8 | Lens Fit Assessment: | when required. |
| 0.8 | Lens Fit Assessment. | Evaluate and grade lens centration, primary gaze movement, upgaze movement and |
| | | tightness (push-up test). |
| | | agnatess (pasit-up test). |
| | | The subject should not proceed to wear the |
| | | lenses if any of the following is observed: |
| | | presence of limbal exposure (appearance) |
| | | of clear cornea) in any gaze |
| | | presence of edge lift |
| | | - |
| | | • presence of unacceptable movement |
| | | (excessive or insufficient) in <u>all three</u> |
| | | movement categories (primary gaze, |

| | Unscheduled Visit | |
|---|---|---|
| | | upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| U.9 | Exit Visual Acuity | Record the subject's exit distance and near visual acuity (OD, OS and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |

# 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

# 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- completed all study visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed two consecutive study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

If more than 2 subjects in the investigational soft contact lens group develop serious expected (e.g., definite or probable MK) or unexpected device related adverse events, the study will be suspended. Upon review and consultation with IRB, DMC, and JJV safety review committee, the study may be terminated. This potential stopping rule is established based on our trial involving approximately 200 subjects wearing the investigational soft contact lens for up to 3 years with an assumed MK rate that is below 0.2% per patient-year. The rate of 0.2% per patient year is the established rate for extended wear lenses in adults, which was requested by the FDA as a criterion for evaluating a contact lens for pediatric use in an FDA response to a

CR-6267, v2.0 JJVC 

pre-IDE submission. To be conservative, 200 independent patient years were used in the calculation. The probability of observing 2 cases or more incidents of MK is 0.061, and 3 cases or more incidents of MK is 0.007 (given an MK rate of 0.2% per patient year).

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJV reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJV, it is determined that it would be unwise to continue at the clinical site.

JJV (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

#### **Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other

unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

# 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events - see definition in Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

• Mild – Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities

- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

# 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the test article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

• Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

None

### 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

CR-6267, v2.0 JJVC 

#### 14. STATISTICAL METHODS

### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type and will be performed separately by completion status (Safety Population or Per-Protocol Population). All analyses will be conducted on per-protocol population (see Section 14.3).

# 14.2. Sample Size Justification

Using the POWER procedure in SAS 9.4, it required at least 59 hyperopic subjects to complete the study to satisfy both primary and secondary hypotheses with overall type I error 0.05 and power no less than 90%. At the end of this section, a summary table of the sample sizes required for each individual hypothesis is provided.

| Primary Hypothesis: | Criteria | # of subjects needed | Power |
|----------------------|------------------|----------------------|-------|
| CLUE Vision | >32 | 19 | 0.9 |
| Secondary Hypothesis | Criteria | # of subjects needed | Power |
| CLUE Vision | Test-Control>=-5 | 59 | 0.9 |

## 14.3. Analysis Populations

### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

# 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 14.5. Primary Analysis

Primary efficacy analysis:

## **CLUE Vision:**

Overall quality of vision scores will be analyzed using a linear mixed model adjusting for baseline values as fixed covariates. The model will include the experimental design factors: sequence of lens wear, period, lens type, time point and interaction between lens and time point as fixed effects. The covariance between residual errors from the same subject across lens wearing periods/time point will be selected based on the finite-sample corrected Akaike's Information Criterion (Keselman et al. 1998)<sup>6</sup>. Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

# **Primary Hypothesis:**

Comparisons will be carried out using 95% confidence intervals constructed of least-square means (LSM) from the linear mixed models of CLUE vision scores for each study population. Statistically superiority will be concluded if the lower limit of the confidence intervals of the test lens are greater than 32 points.

### Secondary Hypothesis:

Comparisons between the test lens and control lens at each time point (1 week and 2 weeks) will be carried out using 95% confidence intervals constructed of least-square means (LSM) differences (Test minus Control) from the linear mixed model. The non-inferiority of the test lens relative to the control will be concluded if the lower confidence limit of LSM difference is above the non-inferiority margin -5. The superiority will be established if the lower confidence limit is above 0.

In all models, the Kenward and Roger method (Kenward and Roger, 1997)<sup>7</sup> will be used for the calculation of the denominator of degrees of freedom.

### 14.6. Secondary Analysis

See section 14.5.

## 14.7. Other Exploratory Analyses

Not Applicable

## 14.8. Interim Analysis

Not Applicable

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJV database manager and sent to JJV for analysis.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 16. DATA MANAGEMENT

### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJV must be contacted and notified in writing within 24 hours.

### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJV. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJV will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJV may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJV and for inspection by local and regulatory authorities.

### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

### 18. ETHICAL AND REGULATORY ASPECTS

### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able

to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)

- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and

regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

## 18.5. Privacy of Personal Data

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the

applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJV.

### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJV management representative prior to study initiation.

JJV reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJV reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Ouery resolution
- Case Report Form signature
- Completion of any follow-up action items

### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: <a href="https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/">https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/</a>
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 6. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. *Communications in Statistics—Simulation and Computation*. 1998;27:591-604.
- 7. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53:983–997.







PRO SPECIFICATIO


2



3








7









1 Final 2018-04-03 PRO SPECIFICATIO 






PRO SPECIFICATIO




17




















28

Protocol 6267



# APPENDIX B: PATIENT INSTRUCTION GUIDE

Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

ACUVUE OASYS® 1-DAY ACUVUE® MOIST MULTIFOCAL 1-DAY ACUVUE® MOIST If vision is acceptable, perform a sittlemp exemination to assess adequate fit contration and movement), if it is acceptable, depense the lenses instructing the patient to what in one week for reseasement (see depending and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at

# TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of sof contact lenses, including lorics, there are some additional steps ansion rules to tollow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUAUE CASYS\* for ASTIG-MATISM contact to rese are that you must determine the stability, repeatability and drift angle of the lens axis so that you can prescribe the correct lens axis for your

### A. How to Determine Lons Cylinder and Axis Orientation

1. Locate the Orientation Marks To help determine the proper orientation of the toric lens, you'll find two primary to hip basishman the proper construction or on the start, but in all we prime marks about it men the liver subgroups representing the vertical position on opposition ands of the later all 8 and 12 to clock (Fig. 1). Bicause of the later basishing system, either mark can special the vertical system. There is no "lipt" and facilities a primit basistated lars. You don't need to view both marks to assess orientation, simply look for the 6 or clock mark as you would with a prism ballated lars.



√ Ingure 1

\*\*Maril read at blemmonocope and a 1 mm or 2 mm parallelephod beam to highlight the marks when the late is filled to the eight three are a number of highlight the marks when the late is filled to the eight three provides produces and modern image profit beam for the ready part down the circle of the marks of the mar

Observe the position and stability of the "bottom" mark, it usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement

Allow the lanses to settle for about 20 minutes with the correct power lanses In place. Walk across the room and have the patient look at you. Assess the in piace. Walk across the noom and have the patient look at you. Assess the patient's reaction to distance vision under these chounterance. Then have the patient look at familier near objects such as a wealth tace or fingernals. Again assess the reaction. As the patient continues to look around the room at both near and delatino objects, observe the reactions. Drily after those vision tests in are completed should the patternt be asked to read print. Evaluate the patt reaction to large print (e.g., hypewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

An initial unfavorable response in the office, while indicative of a guarded prog-nosis, should not immediately rule out a more adorsive trial under the usual conditions in which a patient functions.

4. Adaptation Visually idemanding situations should be avoided during the Initial wearing pe-riod. A patient may at first experience some mild bitured vision, dischasse, has sches, and a feeling of stight imbalance. You should explain the adaptational. symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis

Some patients feel that automobile driving performance may not be optimal Some patients load in that automobile driving performance may not be optimal during the adaption process. This is gentiously five when driving all might. Belone driving a motor varieties, it may be recommended that the patient be a passurgar first to make sure that their death is satisfaction to operating an automobile. During the that search weeks of wear inflamment application is countrig. It may be advisible to the patient to only othe during optimal driving condi-tions. After adaptation and success with these advisition, the patient should be able to drive under other conditions with caution

# D. Other Suggestions

If the monovision factorique may be further improved by having the patient follow the suggestions below

- Have a third contact ions (distance power) to use when critical distance viewing is needed.
- Have a third contact lons (near power) to use when critical near viewing is nearlest
- . Having supplemental spectables to wear over the monovision contact lenses

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still create log out the above the red of the group of the above t swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens. Assessing Retation

Imagine the eye as a clock dial and every hour represents a 30° interest. If the orientative mark of the initial lans stabilizes somewhat left or right of the vertice. oriofization mark of the Initial lans stabilizes somewhat left or right of the vertice position, the final lans will orient on the eye with the same deviation. Ye use use an ask retruile in the sitt lamp or use a line-scribed lens in a spectade hits hame to measure or estimate the "drift angle" of the cylinder axis

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive add to determine the correct cylinder adds. Use the LARS (Left Add, Right Subtrad) method to determine which direction to

### B. How to Determine the Final Lens Power

When the diagnositic lons has its ade aligned in the same meridian as the patient's retractive axis, a spherocylindrical over-retraction may be performed and visual aculty determined. However, in the case of crossed axes, such as are vesse accury obtammined. However, in the case of crossed stoce, such as when the diagnostic lores as is all different from the patients instantive asis, it is not advisable to over-retain because of the difficulty in computing the resultant power. In this gold contact lareas, it is customary to present the text lip ower in the sphere. In the cylinder, however, any lone rotation is visually disturbing to the patient, so its more practical to prescribe as weak a cylinder as possible So, here is how to determine the final iens power.

# For the Sphere:

For the Cylinder:

Adjust the axis by the drift angle using LARS. Choose a cylinder that is < 0.250 from the retractive cylinder.

ions for each eve with an axis as close to 190° as possible. Place the lans on each eye and allow a minimum of 3 minutes to

for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot pass state driv licersing requirements with monovision correction.

 Make use of proper flumination when carrying out visual tasks. Monovision fitting success can be improved by the following succestions

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lans powers if there is trouble with adaptation. Accounte lans power is critical for prosbyopic patients.
- . Emphasize the benefits of clear near vision and straight ahead and upward

e decision to fit a patient with a monovision correction is most appropriately left the Eye Care Professional in conjunction with the patient after carefully consid-

All patients should be supplied with a copy of the PATIENT INSTRUC-TION GUIDE for those lenses. Copies are available for download at www.

# PATIENT MANAGEMENT

# Dispensing Visit

PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULE (DISPOSABLE OR FREQUENT

 Recommend an appropriate cleaning and disinfecting system and provide the patient with instructions regarding proper lens care. Chemical or hydrogen perceide distribution is recommended.

# Schedule a billow-up exemination.

 Follow-up care incoassary to ensure continued supposstul contact lons wear? should include routine periodic progress exeminations, management of specific problems, if any, and a review with the patient of the wear schedule, ions replacement schedule, and proper lens care and handling procedures.

- Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis);
- One week from the initial lons dispensing to petient.
- 3. Every three to six months thereafter

It to equilibrate, based on the patient's initial response to the iens. If the iens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'dook position on both eyes, choose the appropriate cylinder as listed previously. If the ions has not yet stabilized, recheck until stable. Horo is the Ry Prosymbort-

O.D. -2.50 -1.25 x 180 O.S. -2.00 -0.75 x 180

# Example 2

O.S. 475-2001/90 20/20 Choose diagrants lenses of -5.00-0.75 x 90 for the right eye and -4.50 -1.75 x 90 for the left eye, the nearest lenses wellstike to the spherical power and exist reacted. Please the lens on each eye and able an infiltram of 3 minutes for it to equilibrate, based on the patient's tritial response to the lane. If the land has not due to attack lock, cocheck curtil stable. The contratton mark on the right has related to them the 6 o'clock position by 10°. The fitting indicates the following:

Right Eye: Componisate the 10" axis drift by adding it to the manifest refraction axis. -3.00 -0.75 x 100

Left Eye

The lars on the left eye shows good contration, movement and a consistent tendency for the mark to diff right by 10° from the 6 o'clock position tendency for the mark to diff right by 10° from the 6 o'clock position tendenty a propose of 4.750, adjust for the vertex distance and roduce the sphere by 0.750 and 10° from the 10° from prescribe the -1.75D cylinder. Compensate for the 10° axis drift by subtract-ing it from the manifest instruction.

Here is the Rx Prescribed: OS -450-175 x 80

If vision is acceptable, perform a still temp examination to assess adequate till (perfuration and movement). If it is acceptable, dispense the foreas in-structing the pellent to return in one week for reassessment [see dispensing and follow up information in PATIENT MANAGEMENT].

Ill patients should be supplied with a copy of the PATIENT INSTRUCTION UIDE for these lenses. Copies are available for download at

E. More frequent or additional follow-up visits may be recommended for ris on an extended wear schedule.

Profundity, at the follow-up visits, lenses should be worn for at least six hours.

If the lenses are being worn for continuous wear, the exemination should be performed as early as possible on the morning billowing overnight wear.

Recommended Procedures for Follow-Up Visits:

1. Solidit and record patient's symptoms, if any, Measure visual abulty monocularly and bimodularly at distance and near with the contact tensor.

Porform an over-refraction at distance and near to check for residual refractive error.

 With the biomicroscope, judge the iens fitting characteristics (as described in the GENEFAL FITTING GUIDELINES) and evaluate the iens surface for deposits and damage.

Following lans removel, examine the comes and conjunctive with the biomi-croscope and fluorescein funiess contraindicated.

 The presence of vertical corneal striae in the posterior central corner or corneal neovesoulistization is indicative of exceptive corneal eden The presence of corneal staining ancifor limbal-conjunctive hyperemia.

can be indicative of an unclean liens, a reaction to solution preservatives, excessive lens wear, and/or a poorly fitting lens. Papiliary conjunctival changes may be indicative of an unclean and/or damaged lens.

Periodically perform karatometry and spectacle retractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

# WEARING SCHEDULE

Patients land to overwear the lanses initially. The Eve Care Professional should research and as ownersed and interest treate, in e. §ia Cata Protessorial should emphasize the importance of shadning to the hills insulamen wavering should. Maximum wavering time should be determined by the Eye Care Protessorial base upon the patients physiological eye condition, because inclividual response to contact larreas varies.

# MULTIFOCAL FITTING GUIDELINES

c Noods Assessment & Patient Educa

Multiflocal contact lenses may produce compromise to vision under certain directions and the patient should understand that they might not find the vision acceptable in specific situations (i.e., reading a menu in a dim restaura vision acceptable in specifying containing a more in a clim relation of white planting in instripting containing, with previous p

- 2. driving automobiles (e.g., driving at right). Patients who gannot pass their ver's license requirements with these lonses should be advised to with this correction, OR may require that additional over-correction.

hose lanses are not recommended for patients who have -1,000 or greater If refractive cylinder as this level of uncorrected cylinder may lead to additions

These lenses are available in the following ADD powers

. Lans "LOW" = "low" maar ADO lans (Max +1.25 ADO)

. Lans "MID" = "medium" near ADD lens (Max +1.75 ADD) Lans "HGH" = "high" near ADD lons (Max +2.50 ADD)

# B. Fitting Instructions

1. Determine the following:

- Eye dominance (the methods described in MONOVISION FITTING GUIDE-LINES may be used)
- Spinarical equivalent distance prescription (vertex corrects rounded to less minus if between powers)

# 2. Select the initial trial lens as follows:

 For each eye select the trial lens distance power that is closest to the petiont's distance sphortcal equivalent.

The maximum successful waaring time for those lonses is:

| 55 | |
|-------------|-------------------|
| DAY | HOURS |
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waiting hours |

For Extended Wear-It is recommended that the contact lans wasner first be evaluated on a daily wear schedule. If successful, then a gradual introduction of extended wear can be followed as determined by the prescribing Eye Care Professional.

These lanses have been approved for extended wear up to 6 nights/7 days of continuous wear. Not all patients can achieve the maximum wear time. For Therapeutic lons wear, close supervision by the Eve Care Professional is

For immerposes or war, occasing presenting its processing the individual in an increasing the financial mass can be worn for adminded wear for up to 8 nights/7 days of continuous wear. The Eye Care Protessional should determine the appropriate washing time and provide specific instructions to the peakent regarding lars care, insention, and removal.

# REPLACEMENT SCHEDULE

When prescribed for daily wear (frequent replacement), it is recommended that the loneas be discarded and replaced with a new lons every 2 weeks. However, the Eye Care Protessional is encouraged to determine an appropriate replacement schedule based upon the response of the patient.

For Lenses Prescribed for Disposable Weat: What presents but to deposite lever, by the opposition where What presents but to deposite lever, by the opposition of sold due to debt-mitted by the light care followed by the presents the but yet and the constraints, as well as the practificative begathers and official judgment. Once smowed, it is accommended that the law is running out of the eye for a portion of need of contraint or larger and the deceased in accordance with the presentable wearing schools. The light Care Polisopiral should countrie to the patient during the early single of destinated weer.

# . Select the near power of the lens based on the patient's ADD range as

ADD: +0.75 to +1.25 use a "LOW" near ADD lens on each eye ADD: +1.50 to +1.75 use a "MID" near ADD lens on each aw

ADD: +2.00 to +2.50 use a "HGH" near ADD lens on each eye 3. Allow the lone to gettle for a minimum 10 minutes

# 4. Assess distance and near vision binocularly and monocularly.

- Make adjustments in power as necessary (see Multiboal Troubleshooting below). The use of hand-held trial lenses is recommended. If distance and near vision are acceptable, perform a stit tamp exemination to assess adequate fit (contration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see disponsing and follow-up information in PATIENT MANAGEMENT)

onaccoptation near vision:

Colorismin the amount of additional plus, or less minus, over one or both eyes that is acceptable, white checking the effect on distance and near vision. If vision is still not acceptable, change the non-dominant eye to the next highest ACD power.

Unacceptable Distance Vision: Determine the amount of additional minus, or less plus, over one or both eyes Leasmine the amount of adultional minus, or less plus, over one or both of the file acceptable while checking the effect or defance and near vision. If it vision is still not acceptable, change the dominant eye to the next lowest AC power. If the patient is wearing two low ACD lenses, change the dominant eye to a sphero lars with a power equal to the spherical equivalent distance.

inacceptable Distance and Near Vision: letermine the amount of additional plus and/or minus over one or both eyes nat is acceptable while checking the effect on distance and near vision. If and is acceptable what a leading in a check of classified and had vision. If a additional plus and/for minus is not required, change the lans power in the dom frant eye to the next highest ADD power, if applicable.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at

# LENS CARE DIRECTIONS

should recommend an appropriate care system tallored to the patient's individual

ooting and storage, refer to the Patient Instruction Guide for these lenses re available for download at www.aouvus.com.

The Eye Care Professional should review with the patient, lens care directions for cleaning, distributing and storing, including both basic lens care information and specific instructions on the lens care realmen recommended for the patient.

For Lenses Prescribed for Disposable Wear:

# when they are removed and have replacement lenses or spectratics available. Lanses should only be cleaned, rinsed, and disinfected on an emergency bas when replacement lenses or spectracies are not available.

Care for Sticking (Non-Moving) Lenses

The patient should be informed that if chemicals of any kind (household products, gardening solutions, aboratory chamicals, etc.) are spisarbed into the eyes, the pa-tient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CAME PROFESSIONAL, OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY

# MONOVISION FITTING GUIDELINES

Docupational and environmental visual demands should be conside correction. Monovision contact ions wear may not be optimal for activities such

driving automobiles (e.g., driving at night). Petents who cannot pass thair state driver's license requirements with monovision correction should be advised to not drive with this correction, OR may require that additional

ONE continuous segments with a segment of the property of the with the vector produce in visually ordaining in proformants (u.g., heating a menu in a dim restaurant, driving at night in rainyfloggy conditions, etc.). During the fitting process, it is necessary for the patient to rea pward gaze that monovision contact lonses provide.

# B. Eye Selection

1. Ocular Preference Determination Methods Method 1: Determine which eye is the "sighting eye." Have the patient p to an object at the far end of the room. Cover one eye. If the Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-hald this lane equal to the spectate near ADD in fort of one aye and then the other while the distance extractive error connection is in place for both eyes. Determine whether the potent functions best with the near ADD ions over the right or left eve.

 Retractive Error Method
 For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near. 3 Visual Domando Mothod

value terminates wearded.
 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lons on the left eye.

### C. Special Fitting Characteristics

. Unilateral Lens Correction

There are obcurrestances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may only require a distance lons.

Example: A presbyopic emmetropic patient who requires a +1.750 ADD would have a +1.750 lans on the near eye and the other eye laft without a lans. A presbyopic patient requiring a +1.500 ADO who is -2.500 myopic in the right eye and -1.500 myopic in the laft eye may have the right eye corrected for detance and the laft uncorrected for near.

2. Near ADD Delemination

Aways prescribe the lars power for the near eye that provides optic
acutly at the midpoint of the petients habitual reading distance. However than one power provides optimal reading participance, prescribed to the petients of the petients of the petients.

# least plus (most minus) of the powers.

3. Itial Lane Fitting
A Itial Stane Fitting
A Itial Stane Fitting
A Itial Stane Fitting is parformed in the office to allow the patient to experience monowholen connoction. Lareas are fit according to the GENERAL FITTING
GUIDELINES for bease curve existed on in this Packago Insart.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD, With that lenses of the proper power in place, observe the reaction to this mode of correction

IMPORTANT: Please read carefully and keen this.

This Package Insert and Fitting Guide is intended for the Eve lessional, but should be made available to pat

the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at WWW SCHNIEG COM



ACUVUE OASYS® Brand Contact Lenses

ACUVUE OASYS® Brand Contact Lenses for ASTIGMATISM

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily and Extended Wear

R(04) GAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

Each storile ions is supplied in a foll-sealed plastic package containing buffered saline solution with methyl ether collulose. The plastic package is marked with tribution.

 ACUVUE CASYS\*: base curve, power, diameter, lot number, and expiration For complete information or

### ACUVUE OASYS\* for ASTIGMATISM: base ourve, power, diameter, cylinder, axis, lot number, and expiration date ACUVUE OASYS\* for PRESBYOPIA: base curve, power, diameter, ADD, For Lonses Prescribed for Frequent Replacement Wear

The Eye Care Professional should review with patients that no cleaning or disinfac-tion is needed with disposable lanses. Patients should always dispose of lanses

Care for a Dried Out (Dehydrated) Lene

If the frequent replacement lans is off the eye and exposed to air from 30 minutes to 1 frour or more, its surface will become dry and gradually become non-wetting, this should occur, discard the lans and use a new one.

If the lans sticks (stops moving), the patient should be instructed to apply a it in an a some pulpe moving, in a paint include in institution apply at test drops of the recommendate fundating or reweiting solution directly to the eye and well until the lens begins to move heely on the eye below removing it. If it more-movement of the lens continues after a tex minutes, the patient should immediately contact the Eye Care Professional.

EMERGENCIES

Monovision Needs Assessment MONOVARION NOSCE, viewnecement For a good prograsis, the patient should have adequately corrected dista and naar visual acutly in each eye. The amblyopic patient or the patient significant astignation (greater than 1,000) in one eye may not be a good candidate for monovision correction with these lonses.

# visually demanding situations such as operating potentially dange machinery or performing other potentially hazardous activities; any

HOW SUPPLIED

REPORTING OF ADVERSE REACTIONS

All sofous adverse congresses and adverse reactions observed in patients was

Jacksonville, FL 32258

petent is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

upon request. The Eve Care Professional should provide the patient with



ACUVUE OASYS® Brand Contact Lenses for PRESBYOPIA

CR-6267, v2.0 JJVC 

# SYMBOLS KEY

The following symbols may appear on the label or carton-

| | 3,7,4,7 |
|---|---|
| SYMBOL | DEFINITION |
| ŒΙΔ | Consult Instructions for Use |
| - | Manufactured by or in |
| ~ | Date of Manufacture |
| <u> </u> | Use By Date (expiration date) |
| 101 | Batch Code |
| VIIII. | Startie Using Steem or Dry Heat |
| DIA | Diamotor |
| BC | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylindar |
| AXIS | Axis |
| MAX ADO | Near ADD |
| LOW | "Low" Near ADD |
| MID | "Modium" Near ADD |
| HEH | "High" Noar ADD |
| 9686 | Quality System Certification Symbol |
| and Process | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| $F_{X} \cap I_{\ell}$ | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| 9 | Lans Orientation Correct |
| ¥ | Lans Orientation Incorrect (Lans Inside Out) |

"Topping-Off" is the addition of trash solution to solution that has been sitting

# Discard Date on Multi-Purpose Solution Bottle

- Discard any remaining solution after the recommended time period indicated on the bottle of multi-purpose solution used for disinfecting and scaking the contact lenses.
- The Discard Date refers to the time that the patient can safety use contact lens care product after the bottle has been opened. It is not the same as the expiration date, which is the lest date that the product is still effective before it is opened.

Using multi-purpose solution beyond the discard date could result in contemi-nation of the solution and can lead to severe infection, vision loss, or blindness. To avoid contamination, DO NOT touch tip of container to any surface.
Replace cap after using.

- To avoid contaminating the solution, DO NOT transfer to other bottles or

# Instructions for Use

To adequately distribut the lonses, the patient should rub and rinse the lonses according to the recommended lens rubbing and rinsing times in the labeling of the multi-purpose solution WARNING:

- Rub and rinso lonses for the recommended amount of time to help preven
- serrous eye intersors.

  Never use water, saline solution, or reweiting drops to disinfact the lense.

  These solutions will not disinfact the lenses. Not using the recommender disinfaction can lead to severe infaction, vision loss, or billindrass.

# Instructions for Use

- Emply and clean contact lens cases with digital rubbing using fissh, sterile disinfecting solutions/contact lens cleaner. Never use water. Cleaning shoul be followed by rinsing with trash, sterile distributing solutions (hever use water) and wiping the lans cases with heath, clean tissue is recommended. Never air dry or recep the lans case lids after use without any additional cleaning methods. If air drying, be sure that no residual solution remains in the case before allowing it to air dry.
- Replace the lens case according to the directions provided by the Eye Care Professional or the manufacturar's labeling that accompanies the case.

# DESCRIPTION

The ACUNUE CASYS® Brand Contact Lanses, the ACUNUE CASYS® Brand Contact Lanses for ASTIGMATISM, and the ACUNUE CASYS® Brand Contact Lanses or PRESERYOR have soft (hydrophilic) contact lanses switched as sphartos), torto, or multipool lanses and include HYDRACLEAR® PLUS Technology. The lanses are made of a silicone hydrogal material containing an informal wetting agent with visibility timied UV absorbing monomer.

These lenses are tinled blue using Readthy Blue Dye #4 to make the lenses more visible for handling. A benuotriazale UV absorbing monomer is used to block UV

The transmittance characteristics are less than 1% in the UVB rance of 290 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire

#### Lons Proportios:

 Specific Gravity (calculated): 0.98 – 1.12 Retactive Index 85% minimun • Light Transmittance . Surface Character Hydrophilo Water Content:

METHOD WALUE 103 x 10 " (cm²/sac) (mi Oymi x mm Hg) @ 35°C Fatt (boundary corrected, edge corrected) 122 x 10" (cm²/sac) (mi O,/mi x mm Hg) @ 35°C

# Lons Paramotors:

. Diameter Range: 12.0 mm to 15.0 mm Base Curve Range: 7.85 mm to 10.00 mm Daily Waar: -20,000 to +20,000 Multitocal ADD Power Range:

Extended Wear: -20,000 to +14,000 +0.250 to +4.000 2 E7 to 1007

. Cylindar Power Range: Contact lons cases can be a source of bacterial growth

WARNING-WARRINGS:

Do not store lerses or rinse lons cases with water or any non-startle solution.

Only tests multi-purpose solution should be used to prevent contamination of
the lenses or lons case. Use of non-startle solution can lead to severe infection
video loss, or bindhese.

# PRECAUTIONS

 Due to the small number of patients arrolled in dinical investigation of lons Out to the small number of platents enrolled in office interestination of inter-en, all effective powers, design configurations, or interpretations resides in the lens material sea not evaluated in significant numbers. Consequently, when selecting an exproprise lare noteging and personations, the tips Core Professional should consider all characteristics of the lares that can affect lens performance and coular health, including ongigan permastility, worldabil-by, certifial and poliphical thickness, and optic zero demater.

harators, the continuing ocular health of the patient and lens performs on the eye should be carefully monitored by the prescribing Eye Care

- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual soutly for either far or near vision Vexual requirements vary with the individual and should be considered who salecting the most appropriate type of lens for each patient.
- ascein, a yollow dye, should not be used while the lanses are o the eyes. The lonses absorb this dije and become discolored, Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lonses immed-staly if the eyes become red or initiated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precaution

- . DO NOT use if the starfe blister package is opened or damaged.

# AVAILABLE LENS PARAMETERS

The ACUVUE OASYS® Brand Contact Lenses are hemispherical shells of the following dimensions

Confor Thickness Minus Lans - varies with power (e.g. -4.000: 0.070 mm) Plus Lens - varies with power (e.g. +4.000: 0.168 mm)

-0.500 to -6.000 (in 0.250 increment: -6.500 to -12.000 (in 0.500 incremen

The ACLIM IF CASYS® Report Contact Lensus for ASTIGMATISM are homiling helis of the following dimensions:

Diameter: 14.5 mm

Minus Lans - varies with power (e.g. -4.000: 0.080 mm Plus Lens - varies with power (e.g. +4.000: 0.172 mm) 8.6 mm Base Curve:

piano to -6.000 (in 0.250 increments) -6.500 to -9.000 (in 0.500 increments) +0.250 to +6.000 (in 0.250 increments Cylinder: -0.750, -1.250, -1.750, -2.250, -2.750 Axis: 10" to 180" (in 10" increments)

The ACUVUE OASYS® Brand Contact Lanses for PRESBYOPIA are hemispherical shalls of the following dimensions:

#### Diameter: 14.3 mm

Base Curve: 8.4 mm

-9,000 to +6,000 (n.0.250 increments) ADD Powers: +1.25 (LOW), +1.75 (MID), +2.50 (HGH)

- DO NOT touch contact lenses with the fingers or hands if the hands are not tree of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient Instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- Always handle lorses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lanses from the lens containings specifically indicated for that use. Side the lens up the side of the bowl until it is free of the container.
- . Do not touch the lens with fingernalis.

Colons appared in processing the the Therapolatic use of these intress. Color medications used during feathers with a bandage into should be colory medications used during feathers with a bandage into should be colory from the color of the color of the color of the color of the only fine Care Proteotical will next and smooth the larrace. In these colors, plant and the color of the color of the band the feathers of colors.

# Lons Wearing Procautions:

- The harm stoke jetops moving on the eye, billow the recommended directors in 'Care for Bibling (Non-Moving) Lanses'. The lans should mov-healy on the eye for the continued health of the eye. If non-movement of the lars continues, it is polation is houst be instructed to immediately consult his or her Eye Care Protessional.
- Never wear lenses beyond the period recommended by the Eye Care Protessional.
- lonsias. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as heir spray, are used while wearing lenses, exercise caution and leep eyes closed until the spray has settled.
- Avoid all harmful or inflating vapors and furnes while wearing lenses.
- Different solutions cannot always be used together and not all solutions are sate for use with all lenses. Use only recommended solutions.
- Never use solutions recommended for conventional hard contact lenses

# TRANSMITTANCE CURVE



. Larren, S., Radard Energy and the Eye, MacMiller, New York, 1980, p.58, figure 2-21 L Waster, M., Hitchire, V.M., Optical Radation and Vasal Health, CRO Press, Socia Ration, Rorida.

NARNING: UV absorbing contact lenses are NOT substitutes for protein tive UV absorbing eyewear, such as UV absorbing geggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

# ACTIONS

retracting medium to locus light rays on the retine. When hydrated and placed or the comes for therapeutic use, the contact lens acts as a bandage to protect the

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions jailtude, geography, cloud cover) an pursonal factors (axtent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful ÚV radiation

- specifically indicated on product labeling for use in both heat and chemical
- . Always use fresh, unexpired lens care solutions and lenses Do not change solution without consulting with your Eye Care Professions
- Aways follow directions in the package inserts for the use of contact lens
- Use only a chemical (not heat) lors care system. Use of a heat (thermal) care system can damage these lorses. Starile unpreserved solutions, when used, should be discarded after the
- time specified in the directors. Do not use salvs or anything other than the recommended solutions for lubricating or writing lanses.
- Alvegia kopit halvesse completally immersed in the secommended storage solution when the larges completally immersed in the secommended storage solution when the industrial kind in the second plant of the con-dying will notice the ability of the kines authors to have that to a webtiast status. Follow the larse care directions in "Case For A Dried Out [Dehydrated] Lens" flores surbox door boomer defend out.

# Other Topics to Discuss with Patients-

- Aways contact the Eye Care Professional before using any medicine in the exes.
- Contain medications, such as antihistamines, deconquistants, diuretics, Cortain medications, such as artifistatiminas, decongraptine, duratios, muscle insideratis, languillaris, and finesa for motion addresses may cause dryness of the eye, incleased lane sewerness, or bitumed vision. Should is conditions each grouper remodel measures should be prescribed. Deposit participation of the several proper strends measures should be prescribed. Deposit indicated for use with each condition the use of barriorary discontinuation of contact irans were white such medication is being used.
- One contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned
- ng heath or the patients wyw. Immanded blow-up schedule.

# Who Should Know That the Patient is Wearing Contact Lenses'

- . Patients should inform all doctors (Health Care Professionals) about being a contact lons weerer.
- Patients should always inform their employer of being a contact lons wearer Some jobs may require use of eye profection equipment or may require that the patient not wear combact lonses.

# INDICATIONS (USES)

The ACLMUE CASYS® Brand Contact Lons is indicated for the ontical of

The ACLIMUE CASYS® Brand Contact Lons for ASTIGMATISM is indicated for the plical comaction of visual aculty in phakic or aphakic persons with non-diseas yes that are hyperopic or myopic and may have 10.000 or less of astigmatis The ACUMUE CASYS® Brand Contact Lons for PRESBYOPIA is indicated for the optical correction of distance and near vision in presbyopic, phasis or aphasis persons with non-diseased eyes who may have 0.750 or less of astigmatism. These lenses contain a UV Blocker to help protect against transmission of harmful. UV radiation to the comes and into the eye.

Eve Care Professionals may prescribe the lenses either for single-use dispos Eye Case Protessionals may prosorbe the invasis offer for single-use dispos-date was or the participational depolarisms was with clearing indenticion and all diseases the protessional depolarisms of the participation o

nearona:
see Irase are also indicated by thorspoulte use as a bandage lons by the follow-autile and directic coular conditions:
For commal problemtion in list and commal atmormatities such as entropion, technises, beneficially and command arosion. In addition, they are indicated by protection where subtrace or coular shorture maltimative.

- degeneration or paralysis may result in the need to protect the comea from exposure or repeated inflation.
- For comeal pain relief in conditions such as bullous keratopathy, optibalial erosion and abrasion, filamentary keratitis, and post-keratoplasity. For use as a benfor during the healing process of epithelial detects such as chronic epithelial detects, corneal ulcer, neurotrophic and neuroparalytic lenatits, and chemical burns.
- For post surgical conditions where bandage ions use is indicated such as post refractive surgery, lamellar grafts, comeal flaps, and additional ocula

# ADVERSE REACTIONS

- . The eye may burn, sting and/or lich.
- may be less comfort than when the lens was first placed on the eve There may be a feeling of something in the eye (foreign body, scratched
- area. There may be the potential for some lamporary impairment due to purpheral inflitatios, peripheral comeal utions, and comeal eracin. The may be the potential for other physiological observators, such as load generation dealms, comeal movescularization, comeal statings, hipcide trassi administration, this and conjunctivities, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions or redness of
- this eye.

  Poor visual aculty, blurred vision, rainbows or halos around objects, photo-phobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

- tion at least once a cay, may a success

  How do the lenses load on my eyes?

  How do my eyes loak?

  Have I noticed a change in my vision? If the patient reports any problems, he or she should be instructed to IMMEDIATE-LY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new trash lens on the eye.

The patient should be instructed NOT to use a new lons as self-treatment for the The patient should be advised that when any of the above symptoms occur, a serious condition such as infaction, comea disce, necessalistration or this mo-be present. He or she should be instructed to seek immediate protessional lide callon of the protein and prompt treatment to avoid serious eye damage.

surgicus contractors. For situatural stability and protection in plogy back loris fitting where the con-nea and associated surfaces are too impatible to allow the contract rigid gas permacible (PET) pleases to be fit haddlor, the use of the lens can prevent intation and advances in a conditions where there are elevation differences in the hostigraph injection or sear lesson.

ribed for therapeutic use may be worn for daily or extended wearing

# CONTRAINDICATIONS (REASONS NOT TO USE)

- . Acute or subscute inflammation or infection of the anterior chamber of the Any eye disease, injury or abnormality that affects the comea, conjunctive or eyelids
   Severe insufficiency of lacrimal secretion (dry eye)
- Corneal hypoesthesia (reduced corneal sensitivity)
- Any systemic disease that may affect the eye or be exaggerated by wearing contact laneas

- contract stress.

  Allorgh resolutions of coulter surfaces or advises that may be included or energ-genished by wearing contract transe or use of contract trans solutions.

  Outsit inflation due to elargic reactions which may be caused by use of contract trans solutions (a.e., dearing and distributing poliutions, inwesting clopes, inc.), that contact internicate or preservatives (such as marcay or internatives) (a.b.) which came open may develop an adequate an allogic response.
- Any active corneal infection (bacterial, fungal, protozoal or viral)

## WARNINGS

Patients should be advised of the following warnings pertaining to contact

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

# GENERAL FITTING GUIDELINES

# A. Patient Selection: Patients selected to wear these lenses should be chosen based on

- Motivation to wear lanses
   Ability to follow instructions regarding lans wear care
- General health
   Ability to adequately handle and care for the lenses
   Ability to understand the risk and benefits of lens wear

Patients who do not must the above oritoria should not be provided with

contact lenses.

B. Pro-fitting Examination:
Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determine as well as an assessment of their overall ocular, physical, and mental health. Preceding the initial selection of trial contact lenses, a comprehensive coular

Based on this evaluation, If it is determined that the patient is eligible to wear

retractive status and to guide in the selection of the appropriate lens power. Famous to compensate for vertex distance if the retraction is greater than

D. Base Curve Selection (Trial Lons Fitting)
The following this invess should be selected for patients segardises of karatometry readings. However, comed curveture measurements should be performed to establish the patient's beseithe could retain.

 ACLIVLE OASYS\* for ASTIGMATISM- 8.6 mm/14.5 mm ACUVUE OASYS\* for PRESBYOPIA: 8.4 mm/14.3 mm The trial lenses should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

- Loss of Vision

THE DATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESS

- When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious activerse reactions is increased when loneas are worm overright, and that the risk of ulcorative loratitis is greater for extended wear contact lone users than for daily wear users.<sup>3</sup>
- daily week Luens?

  Mallide have shown that contact lens wearors who are smokers have a higher holidance of advance reactions than nonemokers. Problems with contact lenses or lens care products could result in serious highly to the aye. Patients should be calcinated that propor use and care of contact lenses are also are seen products, including lens cases, are assential for the selb-use of those products.
- The overall risk of ulcorative keralitis may be reduced by carefully following directions for lens care, including cleaning the lens case.

New England Journal of Medicine, September 21, 1999; 321 (12), pp. 773-793

### Water Activity

#### Instructions for Use

WARNING:

# loaking and Storing Your Lenses

Instructions for Use Use only hash multi-purpose (contact lans disinfacting) solution each time the

Do not rease or "top off" old solution left in the lares case since solution reuse reduces effective lares disinfaction and could lead to severe infection, vision loss, or blinchess.

Chinas of a Property RT Lone. A property if the red contrained completely cover the comes (i.e., no limbel as possarly, have sufficient movement to provide loar exchange under the contact lars with no brink, and be controlled. The term should move healy when manipulated digitally with his lower list, and then return to its property centered position when released.

Criteria of a Flat Fitting Lons
 A flat fitting lans may exhibit one or more of the following characterists:

A fast training sins may define one or more of the bloowing characteristics; decentration, incomplete contend coverage (i.e., limbel exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be fast fitting, it should not be dispersed to the patient.

3. Otheris of a Steep Fitting Lans.
A steep thing lars may satisfied one or more of the following characteristics: insultant movement with the blink, conjunctived indomission, and soletance when pushing the lars up digitally with the lower list. If the lars is judged to be steep fitting, in should not be depended to the potant.

If the Initial trist beas curve is judged to be fait or steep fitting, the alternate beas curve, if available, should be trial fit and evaluated after the patient has adjusted to the time. The lares fould move heavy when manipulated digitally with lower lid, and then nature to a property contained position when reliaised. If relations 

Example 1

E. Final Lens Power (Spherical)

E. Final Lens Power (Spherical)

E. Final Lens Power (Spherical)

E. Final Lens Power (Spherical) A sprantice over-remarker and/or to previously the sprantial over-remarker is not as an power after the rise till is judged accorptable. The sprantial over-refraction should be combined with the trial lens power to determine the first larse pre-scription. The pollient should separation good visual aculty with the contect larse power unless there is excessive residual antigrations.

| Spherical over-refraction: | -0.250 |
|----------------------------|--------|
| Final lons power: | -2.250 |
| Example 2 | |
| Diagnostic lons- | -2.000 |

CR-6267, v2.0 JJVC 

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Instruction Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



1-DAY ACUVUE® MOIST Brand Contact Lenses

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses

etafilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

# SYMBOLS KEY

The following symbols may appear on the label or packaging:

| SYMBOL | DEFINITION |
|------------|-----------------------------------------------------|
| Ţį | Consult Instructions for Use |
| | Manufacturer |
| سا | Date of Manufacture |
| | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterilized Using Steam Heat |
| 8 | Do Not Re-Use (Single Use) |
| <b>™</b> ✓ | Lens Orientation Correct |
| X X | Lens Orientation Incorrect (Lens Inside Out) |
| C€<br>0086 | Quality System Certification Symbol |
| 0 | Fee Paid for Waste Management |
| EC REP | Authorized Representative in the European Community |

Visit www.acuvue.com/guides for additional information about symbols.

# DESCRIPTION

1-DAY ACUVUE® MOIST Brand Contact Lenses, 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM, and 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are soft (hydrophilic) contact lenses available as spherical, toric, or multifocal lenses, and include LACREON® Technology.

The lens material (etaflicon A) is a copolymer of 2-hydroxyethyl methacrylate and methacrylic acid cross-linked with 1, 1, 1-trimethylol propane trimethacrylate and ethylene glycol dimethacrylate.

The lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. A benzotriazole UV absorbing monomer is used to block UV radiation.

## Lens Properties:

The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 – 1.12

Refractive Index: 1.40

Light Transmittance: 85% minimum
 Surface Character: Hydrophilic
 Water Content: 58%

Oxygen Permeability (D/k):

VALUE METHOD

21.4 x 10 11 (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge corrected)

(ml O,/ml x mm Hg) @ 35°C

28.0 x 10 11 (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-edge corrected)

(ml O,/ml x mm Hg) @ 35°C

# Lens Parameters Ranges:

Diameter (DIA): 12.0 mm to 15.0 mm
 Center Thickness: Varies with power
 Base Curve (BC): 7.85 mm to 10.00 mm
 Spherical Power (D): -20.00D to +20.00D
 Cylinder Power (CYL): -0.25D to -10.00D
 Axis (AXIS): 2.5° to 180°
 ADD Powers: +0.25D to +4.00D

# **AVAILABLE LENS PARAMETERS**

1-DAY ACUVUE® MOIST Brand Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.2 mm

Center Thickness: 0.084 mm to 0.230 mm (varies with power)

Base Curve (BC): 8.5 mm, 9.0 mm

Powers (D): -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments)

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are hemitoric

shells of the following dimensions:

Diameter (DIA): 14.5 mm

Center Thickness: 0.090 mm to 0.189 mm (varies with power)

Base Curve (BC): 8.5 mm

**Powers (D):** +0.00 to -6.00D (in 0.25D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\*

Axis (AXIS): 10° to 180° in 10° increments

\*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°,

100°, 110°, 160°, 170°, 180° axes only

-6.50D to -9.00D (in 0.50D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10°, 20°, 60°, 70°, 80°, 90°, 100°, 110°,

120°, 160°, 170°, 180°

\*-2.25D cylinder is available in 20°, 90°, 160°, 180°

axes only

+0.25D to +4.00D (in 0.25D increments) Cylinders (CYL): -0.75D, -1.25D, -1.75D

Axis (AXIS): 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.3 mm

Center Thickness: 0.084 mm to 0.207 mm (varies with power)

Base Curve (BC): 8.4 mm

**Powers (D):** +6.00D to -9.00D (in 0.25D increments)

Near ADD Powers Low Near ADD (LOW): +1.25D (MAX ADD): Low Near ADD (MID): +1.75D Medium Near ADD (MID): +1.75D

High Near ADD (HGH): +2.50D

4

# TRANSMITTANCE CURVES

1-DAY ACUVUE® MOIST Brand Contact Lenses (etaflicon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



\*The data are representative measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-3.00D lens, 0.084 mm center thickness).

<sup>1</sup> Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21
<sup>2</sup> Waxler, M., Hitchins, V.M., Optical Radiation and Visual Heath, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

# **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

The UV Blocking for these lenses averages 97% in the UVB range of 280 nm to 315 nm and 82% in the UVA range of 316 nm to 380 nm for the entire power range.

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

# INDICATIONS (USES)

1-DAY ACUVUE® MOIST Brand Contact Lenses are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1,000 or less of astiomatism.

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.500 to 3.000 of astigmatism.

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are indicated for daily disposable wear for the optical correction of distance and near vision in presbyopic phakic or aphakic persons with non-diseased eyes who may have 4.00D of ADD power or less and 0.75D or less of astigmatism.

The lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

When prescribed for daily disposable use, no cleaning or disinfection is required. Lenses should be discarded upon removal.

# CONTRAINDICATIONS (REASONS NOT TO USE)

# DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eve.
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
- Severe insufficiency of lacrimal secretion (dry eye).
- Corneal hypoesthesia (reduced corneal sensitivity).

- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions,
- Ocular irritation due to allergic reactions which may be caused by use
  of contact lens solutions (i.e., rewetting drops) that contain chemicals or
  preservatives (such as mercury, Thimerosal, etc.) to which some people
  may develop an allergic response.
- · Any active corneal infection (bacterial, fungal, protozoal, or viral).
- · If eyes become red or irritated.

# **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- Eve Discomfort.
- Excessive Tearing,
- Vision Changes.
- · Loss of Vision,
- Eve Redness, or
- · Other Eye Problems,

# THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- When prescribed for daily wear, patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that when lenses are worn overnight, the risk of ulcerative keratitis is greater than among those who do not wear them overnight.<sup>3</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.

7

 The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

<sup>3</sup>New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

# Specific Instructions for Use and Warnings:

### Water Activity

Instruction for Use

Do not expose contact lenses to water while wearing them.

### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

# **PRECAUTIONS**

# Special Precautions for Eye Care Professionals:

 Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

 Patients who wear these lenses to correct presbyopia using monovision (or modified monovision using 1-DAY ACUVUE® MOIST Brand MULTIFOCAL) may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.

- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

# Handling Precautions:

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- · DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.
- · Do not touch the lens with fingernails.

# Lens Wearing Precautions:

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for Sticking (Non-Moving) Lenses." The lens should move freely on the eye for the continued health of the eye. If nonmovement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.

- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hairspray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.

### Lens Care Precautions:

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

# Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

# Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

# **ADVERSE REACTIONS**

The patient should be informed that the following problems may occur when wearing contact lenses:

- · The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal uicers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- · How do the lenses feel on my eyes?
- · How do my eyes look?
- · Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or irltis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

# **GENERAL FITTING GUIDELINES**

# A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses
- · Ability to follow instructions regarding lens wear
- · General health
- Ability to adequately handle and care for the lenses
- · Ability to understand the risks and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

# B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

# C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D.

## D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

- 1-DAY ACUVUE® MOIST: 8.5 mm/14.2 mm
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: 8.5 mm/14.5 mm
- 1-DAY ACUVUE® MOIST MULTIFOCAL: 8.4 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

# 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

# 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

# 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

# E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

| Example 1 | |
|------------------------------------------------|------------------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | |
| Diagnostic lens: | -2.00D |
| Diagnostic lens:<br>Spherical over-refraction: | -2.00D<br>+0.25D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing 1-DAY ACUVUE® MOIST for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

# A. How to Determine Lens Cylinder and Axis Orientation

## 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.



You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

# 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift," measure or estimate the "drift," then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

### B. Final Lens Power

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

# 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx > 4.00D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq \pm 4.00D$ , vertex compensation is not necessary.

# 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq$  0.50D from the refractive cylinder.

## 3. Case Examples

# Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20

O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

# Example 2

Manifest (spectacle) refraction:

O.D. -3.00D / -1.00D x 90° 20/20

O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

### Right Eve

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx prescribed:

O.D. -3.00D / -0.75D x 100°

# Left Eve

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx prescribed:

O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see

PATIENT MANAGEMENT section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# MULTIFOCAL FITTING GUIDELINES

# A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with 1-DAY ACUVUE® MOIST MULTIFOCAL. Wearing these lenses may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet
  their state driver's license requirements with the 1-DAY ACUVUE® MOIST
  MULTIFOCAL should be advised to not drive with this correction, OR may
  require that additional over-correction be prescribed.

1-DAY ACUVUE® MOIST MULTIFOCAL is not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise. These lenses are available in the following ADD powers:

- Lens "LOW" = low near ADD lens (Max ADD +1.25)
- Lens "MID" = medium near ADD lens (Max ADD +1.75)
- Lens "HGH" = high near ADD lens (Max ADD +2.50)

### R. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D. Determine the spherical equivalent distance prescription for a multifocal patient. Determine the eye dominance using one of the methods below:

- Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.
- Method 2 Determine which eye does not accept added plus power. Place a +1.00D hand-held trial lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes while the patient is viewing the distance visual acuity chart. The eye with the plus over it that the patient notices the greatest reduction in vision is determined to be the dominant eye.

### C. Select the Initial Trial Lens

- For each eye, select the trial lens distance power that is closest to the
  patient's distance spherical equivalent. Remember to compensate for
  vertex distance if the refraction is greater than ±4,00D.
- Select the near power of the lens based on the patients ADD range as follows:
  - ADD: +0.75D to +1.25D use a low near ADD (LOW) lens on each eye
  - ADD: +1.50D to +1.75D use a medium near ADD (MID) lens on each eve
  - ADD: +2.00D to +2.50D use a medium near ADD (MID) on the dominant eye and a high near ADD (HGH) lens on the non-dominant eye
- 3. Allow the lenses to settle for a minimum of 10 minutes.
- 4. Assess distance and near vision binocularly and monocularly.
- Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate, and near.
- Make adjustments in power as necessary based on the distance overrefraction. The use of hand-held trial lenses is recommended. Check the impact on distance and near vision.
- 7. If vision is still unacceptable, make adjustments in power as necessary (see "Multifocal Troubleshooting" below). If distance and near vision are acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

# D. Multifocal Troubleshooting

## **Unacceptable Near Vision**

If it has been determined that no change is required based on the overrefraction, then add +0.25D to the spherical power of the non-dominant eye.

# Unacceptable Distance Vision

If it has been determined that no change is required based on the overrefraction, then make the changes as listed below:

- If the patient is wearing two "LOW" ADD lenses, change the dominant eye to a 1-DAY ACUVUE® MOIST sphere lens with a power equal to the spherical equivalent distance prescription.
- If the patient is wearing two "MID" ADD lenses, change the ADD power in the dominant eve to the "LOW" ADD power.
- If the patient is wearing a "MID" ADD lens in the dominant eye and a "HGH" ADD lens in the non-dominant eye, change the non-dominant eye to a "MID" ADD lens and add +0.25D to the distance power.

## E. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# MONOVISION FITTING GUIDELINES

### A. Patient Selection

## 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet their state driver's license requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual aculty and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dimly lit restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

# **B. Eve Selection**

### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eve. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eve.

Method 2 Determine which eve will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eve and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

# 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

# Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

# Visual Demands Method

Consider the patient's occupation during the eve selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eve on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

# C. Special Fitting Characteristics

### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on both eyes.

### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left eye uncorrected for near.

### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

## 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the **GENERAL FITTING GUIDELINES** for base curve selection described in this Package Insert.

Case history and a standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next, determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted. An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

# D. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision, and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# PATIENT MANAGEMENT

- Follow the accepted standard of care in fitting and following up with your patient, e.g., American Optometric Association standard of care.
- · Schedule the appropriate follow-up examination.
- Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses, which can be found at www.acuvue.com. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

# WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.
The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

#### REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

When disposed of after a single daily use, these lenses may reduce the risk of developing giant papillary conjunctivitis.<sup>4</sup>

When worn as a daily disposable lens, these lenses may provide improved comfort for many patients who experience mild discomfort and itching associated with allergies during contact lens wear, compared to lenses replaced at intervals of greater than 2 weeks.

Clinical research has shown that when worn on a daily disposable basis, these lenses may provide improved comfort for 2 out of 3 patients who reported suffering from discomfort associated with allergies during contact lens wear.

#### LENS CARE DIRECTIONS

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have replacement lenses or spectacles available.

For complete information concerning contact lens handling and care, refer to the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### Care for Sticking (Non-Moving) Lenses

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution

<sup>&</sup>lt;sup>4</sup>The CLAO Journal, July 1999, Volume 25, Number 3

directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should **immediately** consult the Eye Care Professional.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

#### **HOW SUPPLIED**

Each UV-absorbing sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with povidone. The plastic package is marked with the following:

- 1-DAY ACUVUE® MOIST: base curve, power, diameter, lot number, and expiration date
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date
- 1-DAY ACUVUE® MOIST MULTIFOCAL: base curve, power, diameter, ADD power, lot number, and expiration date

#### REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

> Tel: 1-800-843-2020 www.acuvue.com



©Johnson & Johnson Vision Care, Inc. 2017 In Canada: Johnson & Johnson Vision Care division of Johnson & Johnson Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed In USA Revision date: 07/17 Revision number: M-07-17-02

> 1-DAY ACUVUE® MOIST and LACREON® are Trademarks of Johnson & Johnson Vision Care, Inc.

### APPENDIX D: BINOCULAR OVER REFRACTION

# Binocular Over-refraction Technique

- 1. Place trial frame on subject
- 2. Add +1.00 D sphere to OS
- 3. Add + 0.50DS OD and check VA
  - if VA remained unchanged or improved, repeat step 3
  - if VA decreased, add minus until best VA first achieved \*note: add minus for 0.5 seconds to avoid reflex accommodation.
- 4. Record VA
- 5. Change +1.00 D sphere to OD
- 6. Repeat steps 3 and 4

### APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

### **Presbyopic Symptoms Questionnaire**

- 1. Do you notice that you often have to hold things farther away so that you can read them?
- 2. Do you notice that you often have difficulty focusing on near objects (i.e., experiencing blurry vision when looking at things close-up)?
- 3. Do you often have headaches or eyestrain, or feel fatigued, when reading or conducting other near activities?
- 4. Do you often have difficulty reading small or fine prints, such as phone books, medicine bottles or package labels, etc.?
- 5. Do you often have difficulty reading under dim or low light?

#### OCULAR DOMNANCE TEST

#### +1.00 D LENS TEST

- Step 1 Place the subjects best sphero-cylindrical distance refraction in a trial frame.
- Step 2 Have the subject view a BVA line of letters.
- Step 3 With both eyes open alternate a +1.00 D trial lens between the right and left eye and ask the subject to indicate over which eye does the lens cause the line of letters to appear more blurred. The eye that the greatest blur is reported is the distance dominant eye. If the subject indicates that the amount of blur is about the same between the two eyes then record as neither eye dominant.

#### SIGHTING OCULAR DOMINANCE

- Step 1 Ask the subject to extend both arms out and use his/her hands to form a triangle. The subject will be asked to keep both eyes open, and look through the triangle at a small object on the wall (e.g., a light switch or doorknob).
- Step 2 Occlude the subject's left eye, then right eye. While alternating the occluder from the subject's eyes, ask the subject when they see the object.

If the subject sees the object when the left eye is covered, the subject is *right eye* dominant.

If the subject sees the object when the right eye is covered, the subject is *left eye* dominant.

If the subject sees the object with both eyes, the opening between the hands may be too large. Therefore, ask the subject to make a smaller opening and repeat the procedure.

### APPENDIX G: TEST LENS FITTING GUIDE

### **Step 1.**

Choose the first lens based on the best spherical equivalent refraction and ADD power for both eyes. Select the first lens per table 1 below.

Table 1. Initial Lens Selection

| | ADD | | | | | | | |
|--------------|-------|-------|-------|-------|-------|-------|-------|-------|
| | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant Eye | LOW | LOW | LOW | MID | MID | MID | MID | MID |
| Non- | | | | | | | | |
| Dominant Eye | LOW | LOW | LOW | MID | MID | HGH | HGH | HGH |

Assess the subject's vision at distance and near after the lens has settled (10 minutes). If the vision is acceptable continue with the fit assessment and dispensing as per the protocol.

If the vision is not acceptable, ensure that the proper initial lens power was selected by performing a distance over-refraction with +/- 0.25D trial lenses (or flippers) to determine if a change in the initial lens power is required (note: the over-refraction should be performed outside of the phoropter in normal room illumination). Recheck both distance and near vision with the over-refraction in place. If a change in the initial lens power is not required refer to the fitting steps listed below in step 2 (table 2).

### Step 2.

Table 2. Lens change if required. \*

| Distance<br>Complaint | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| ADD | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant<br>Eye | ACUVUE® OASYS® 2-WEEK Sphere | ACUVUE® OASYS® 2-WEEK Sphere | ACUVUE® OASYS® 2-WEEK Sphere | LOW | LOW | MID | MID | MID |
| Non-<br>Dominant<br>Eye | LOW | LOW | LOW | MID | MID | MID<br>+ | MID<br>+ | MID<br>+ |

| Near | | | | | | | | |
|-----------|-------|-------|-------|-------|-------|-------|-------|-------|
| Complaint | | | | | | | | |
| ADD | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant | | | | | | | | |
| Eye | LOW | LOW | LOW | MID | MID | MID | MID | MID |
| Non- | | | | | | | | |
| Dominant | LOW+ | LOW+ | LOW+ | MID+ | MID+ | HGH+ | HGH+ | HGH+ |
| Eye | | | | | | | | |

<sup>\*</sup>Note: a + following the contact lens design indicates to add +0.25 D to the distance contact lens power on the non-dominant eye (see example below).

Example: The subject is a +1.75 ADD and has a near complaint and it is determined a change in lens pairs is needed. Referring to table 2 near complaint section, under the +1.75 ADD it states to keep the dominant eye the same (i.e. MID) and add +0.25D to the non-dominant eye (i.e. MID+).

## Subjects spherical equivalent distance refraction

OD: +2.50

OS: +3.00 (OS non-dominant eye)

#### The new lens chosen should be as follows:

OD: +2.50 MID ADD (i.e. no change)

OS: +3.25 MID ADD

# **Step 3**.

If after the above lens modifications have been attempted and the subject's vision is still not satisfactory, and additional optimizations are allowed by the protocol, lens changes may be attempted, based on the Investigator's clinical experience, to determine if acceptable vision can be achieved.

#### APPENDIX H: CONTROL LENS FITTING GUIDE

### **Step 1.**

Choose the first lens based on the best spherical equivalent refraction and ADD power for both eyes. Select the first lens per table 1 below.

Table 1. Initial Lens Selection

| | ADD | | | | | | | |
|--------------|-------|-------|-------|-------|-------|-------|-------|-------|
| | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant Eye | | | | | | | | |
| | LOW | LOW | LOW | MID | MID | MID | MID | MID |
| Non- | | | | | | | | |
| Dominant Eye | LOW | LOW | LOW | MID | MID | HGH | HGH | HGH |

Assess the subject's vision at distance and near after the lens has settled (10 minutes). If the vision is acceptable continue with the fit assessment and dispensing as per the protocol.

If the vision is not acceptable, ensure that the proper initial lens power was selected by performing a distance over-refraction with +/- 0.25D trial lenses (or flippers) to determine if a change in the initial lens power is required (note: the over-refraction should be performed outside of the phoropter in normal room illumination). Recheck both distance and near vision with the over-refraction in place. If a change in the initial lens power is not required refer to the fitting steps listed below in step 2 (table 2).

### Step 2.

Table 2. Lens change if required. \*

| Distance<br>Complaint | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| ADD | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant<br>Eye | 1-Day<br>ACUVUE®<br>Moist | 1-Day<br>ACUVUE®<br>Moist | 1-Day<br>ACUVUE®<br>Moist | LOW | LOW | MID | MID | MID |
| Non-<br>Dominant<br>Eye | LOW | LOW | LOW | MID | MID | MID<br>+ | MID<br>+ | MID<br>+ |

| Near | | | | | | | | |
|-----------|-------|-------|-------|-------|-------|-------|-------|-------|
| Complaint | | | | | | | | |
| ADD | +0.75 | +1.00 | +1.25 | +1.50 | +1.75 | +2.00 | +2.25 | +2.50 |
| Dominant | | | | | | | | |
| Eye | LOW | LOW | LOW | MID | MID | MID | MID | MID |
| Non- | | | | | | | | |
| Dominant | LOW+ | LOW+ | LOW+ | MID+ | MID+ | HGH+ | HGH+ | HGH+ |
| Eye | | | | | | | | |

<sup>\*</sup>Note: a + following the contact lens design indicates to add +0.25 D to the distance contact lens power on the non-dominant eye (see example below).

Example: The subject is a +1.75 ADD and has a near complaint and it is determined a change in lens pairs is needed. Referring to table 2 near complaint section, under the +1.75 ADD it states to keep the dominant eye the same (i.e. MID) and add +0.25D to the non-dominant eye (i.e. MID+).

## Subjects spherical equivalent distance refraction

OD: -2.50

OS: -3.00 (OS non-dominant eye)

#### The new lens chosen should be as follows:

OD: -2.50 MID ADD (i.e. no change)

OS: -2.75 MID ADD

#### Step 3.

If after the above lens modifications have been attempted and the subject's vision is still not satisfactory, and additional optimizations are allowed by the protocol, lens changes may be attempted based on the Investigator's clinical experience, to determine if acceptable vision can be achieved.

# **APPENDIX I:**

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
   EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
   DETERMINATION OF NEAR ADD
   NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
   LENS FITTING CHARACTERISTICS
   SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION
  TESTING

# LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS



rage ror


















CR-6267, v2.0









# **DETERMINATION OF NEAR ADDITION**






























# LENS FITTING CHARACTERISTICS














## SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS




# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















### **BIOMICROSCOPY SCALE**
















### KERATOMETRY PROCEDURE




### DISTANCE AND NEAR VISUAL ACUITY EVALUATION












# DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE









#### VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION















#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

CR-6267 Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population

Version and Date: 2.0 Amendment 1 22 June 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| - | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |